CLINICAL TRIAL: NCT03980483
Title: A 52-week, Phase 3, Multicentre, Randomised, Double Blind, Efficacy and Safety Study Comparing GSK3196165 With Placebo and With Tofacitinib, in Combination With Methotrexate in Participants With Moderately to Severely Active Rheumatoid Arthritis Who Have an Inadequate Response to Methotrexate
Brief Title: Efficacy and Safety of GSK3196165 Versus Placebo and Tofacitinib in Participants With Moderately to Severely Active Rheumatoid Arthritis Who Have an Inadequate Response to Methotrexate
Acronym: contRAst 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201790
Record Dates: First submitted 2019-05-15; First posted 2019-06-10 (Actual); Results first posted 2023-10-25 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Arthritis, Rheumatoid
Keywords: Rheumatoid arthritis; GSK3196165; Otilimab; Tofacitinib; Methotrexate; Placebo
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Otilimab; tofacitinib

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of six intervention arms in ratio of 6:6:3:1:1:1.
Who Masked: Participant, Investigator
Masking Description: Double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- GSK3196165 90mg + MTX (Experimental): Participants received GSK3196165 90 mg subcutaneous (SC) injection once weekly for 52 weeks in combination with methotrexate (MTX).
  Interventions: Biological: GSK3196165 (Otilimab)
- GSK3196165 150mg + MTX (Experimental): Participants received GSK3196165 150 mg subcutaneous (SC) injection once weekly for 52 weeks in combination with MTX.
  Interventions: Biological: GSK3196165 (Otilimab)
- Tofacitinib 5mg + MTX (Active Comparator): Participants received Tofacitinib 5mg capsule, orally, twice daily (BID) in combination with MTX plus placebo injection weekly to maintain the blind for 52 weeks.
  Interventions: Drug: Tofacitinib 5 mg
- Placebo + MTX and GSK3196165 90mg + MTX (Placebo Comparator): Participants received Placebo weekly SC injection in combination with MTX for 12 weeks. At Week 12, participants were switched from placebo to GSK3196165 90 mg, SC injection, once weekly in combination with MTX until Week 52.
  Interventions: Biological: GSK3196165 (Otilimab); Drug: Placebo
- Placebo + MTX and GSK3196165 150mg + MTX (Placebo Comparator): Participants received Placebo weekly SC injection in combination with MTX for 12 weeks. At Week 12, participants were switched from placebo to GSK3196165 150 mg, SC injection, once weekly in combination with MTX until Week 52.
  Interventions: Biological: GSK3196165 (Otilimab); Drug: Placebo
- Placebo + MTX and Tofacitinib 5mg + MTX (Placebo Comparator): Participants received Placebo capsule weekly in combination with MTX for 12 weeks. At Week 12, participants were switched from placebo capsule to Tofacitinib 5mg, capsule, orally, BID in combination with MTX plus placebo injection to maintain the blind for 52 weeks.
  Interventions: Drug: Tofacitinib 5 mg; Drug: Placebo

INTERVENTIONS:
Biological: GSK3196165 (Otilimab) — GSK3196165 solution in vial/pre-filled syringe (PFS) to be administered SC.
  Arms: GSK3196165 150mg + MTX; GSK3196165 90mg + MTX; Placebo + MTX and GSK3196165 150mg + MTX; Placebo + MTX and GSK3196165 90mg + MTX
Drug: Tofacitinib 5 mg — Tofacitinib cap (over encapsulated 5mg tablet) to be administered orally.
  Arms: Placebo + MTX and Tofacitinib 5mg + MTX; Tofacitinib 5mg + MTX
Drug: Placebo — Placebo sterile 0.9 percentage (%) weight by volume (w/v) sodium chloride solution in vial/pre-filled syringe (PFS) to be administered SC.
  Arms: Placebo + MTX and GSK3196165 150mg + MTX; Placebo + MTX and GSK3196165 90mg + MTX
Drug: Placebo — Placebo cap (containing lactose) to be administered orally.
  Arms: Placebo + MTX and Tofacitinib 5mg + MTX

SUMMARY:
This study [contRAst 1 (201790: NCT03980483)] is a phase 3, randomized, multicenter, double blind study to assess the safety and efficacy of GSK3196165, in combination with methotrexate (MTX), for the treatment of adult participants with moderate to severe active rheumatoid arthritis (RA) who have had an inadequate response to MTX. The study will consist of a screening phase of up to 6 weeks followed by a 52-week treatment phase in which participants will be randomized in a ratio of 6:6:3:1:1:1 to receive GSK3196165 150 milligrams (mg) subcutaneous (SC) weekly, GSK3196165 90 mg SC weekly, tofacitinib capsules (cap) 5 mg twice a day or placebo (three arms, each placebo arm will have 12 weeks placebo followed by 40 weeks active treatment) respectively, all in combination with MTX. Participants who, in investigator's judgement will benefit from extended treatment with GSK3196165, may be included in the long-term extension study [contRAst X (209564: NCT04333147)]. For those participants who do not continue into the long term-extension study, there will be an 8 week safety follow-up visit following the treatment phase.

ELIGIBILITY:
Key inclusion criteria

* >=18 years of age
* Has had RA for >=6 months and was not diagnosed before 16 years of age
* Has active disease, as defined by having both:*

  * >=6/68 tender/painful joint count (TJC), and
  * >=6/66 swollen joint count (SJC)
* Has at least 1 bone erosion present on hand/wrist or foot radiographs
* Has had an inadequate response to MTX, despite currently taking MTX 15-25 mg/week** oral or injected

  * If surgical treatment of a joint has been performed, that joint cannot be counted in the TJC or SJC.

    * A lower dose of 7.5 mg/week is acceptable if reduced for reasons of intolerance to MTX or per local requirement.

Key exclusion criteria

* Has had any active and/or recurrent infections (excluding recurrent fungal infections of the nail bed) or has required management of acute or chronic infections.
* Has received prior treatment with an antagonist of GM-CSF or its receptor or Janus kinase (JAK) inhibitors (either experimental or approved)
* Has received prior treatment with a biologic Disease-modifying antirheumatic drug (DMARD) which has been discontinued due to an inadequate response.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1537 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2022-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (58):
- China (5):
  - GSK Investigational Site, Bengbu, Anhui
  - GSK Investigational Site, Pingxiang, Jiangxi
  - GSK Investigational Site, Changchun, Jilin
  - GSK Investigational Site, Chengdu, Sichuan
  - GSK Investigational Site, Shanghai
- Hungary (7):
  - GSK Investigational Site, Baja
  - GSK Investigational Site, Balatonfüred
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Kistarcsa
  - GSK Investigational Site, Szentes
  - GSK Investigational Site, Székesfehérvár
  - GSK Investigational Site, Veszprém
- India (15):
  - GSK Investigational Site, Ahmedabad
  - GSK Investigational Site, Banglore
  - GSK Investigational Site, Belagavi
  - GSK Investigational Site, Hubli
  - GSK Investigational Site, Hyderabad
  - GSK Investigational Site, Jaipur
  - GSK Investigational Site, Kolkata
  - GSK Investigational Site, Nagpur
  - GSK Investigational Site, Nashik
  - GSK Investigational Site, New Delhi
  - GSK Investigational Site, Pimpri-Chinchwad
  - GSK Investigational Site, Pune
  - GSK Investigational Site, Rajkot
  - GSK Investigational Site, Surat
  - GSK Investigational Site, Vadodara
- GSK Investigational Site, Verona, Veneto, Italy
- Malaysia (4):
  - GSK Investigational Site, Klang
  - GSK Investigational Site, Kuala Lumpur
  - GSK Investigational Site, Seremban, Negeri Sembilan
  - GSK Investigational Site, Sibu
- Poland (18):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Częstochowa
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Gdynia
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Nowa Sól
  - GSK Investigational Site, Olsztyn
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Sochaczew
  - GSK Investigational Site, Staszów
  - GSK Investigational Site, Torun
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
  - GSK Investigational Site, Zamość
- GSK Investigational Site, Moscow, Russia
- GSK Investigational Site, Belgrade, Serbia
- Spain (3):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Santiago de Compostela
- United Kingdom (3):
  - GSK Investigational Site, Romford, Essex
  - GSK Investigational Site, Northwood, Middlesex
  - GSK Investigational Site, Kenilworth, Warwickshire

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Background] Fleischmann RM, van der Heijde D, Strand V, Atsumi T, McInnes IB, Takeuchi T, Taylor PC, Bracher M, Brooks D, Davies J, Goode C, Gupta A, Mukherjee S, O'Shea C, Saurigny D, Schifano LA, Shelton C, Smith JE, Wang M, Wang R, Watts S, Weinblatt ME. Anti-GM-CSF otilimab versus tofacitinib or placebo in patients with active rheumatoid arthritis and an inadequate response to conventional or biologic DMARDs: two phase 3 randomised trials (contRAst 1 and contRAst 2). Ann Rheum Dis. 2023 Dec;82(12):1516-1526. doi: 10.1136/ard-2023-224482. Epub 2023 Sep 12. PMID 37699654
- See also: 209564 contRAst X NCT04333147 — https://clinicaltrials.gov/ct2/show/NCT04333147?term=209564&draw=2&rank=1

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized in ratio of 6:6:3:1:1:1 to GSK3196165 90 milligram (mg):GSK3196165 150mg:Tofacitinib 5mg:Placebo:Placebo:Placebo. At Week 12, participants randomized to one of the three placebo arms switched to active intervention arms (either GSK3196165 150mg, GSK3196165 90mg or Tofacitinib 5mg BID) receiving active intervention for 40 weeks. Participants randomized to GSK3196165 90mg, GSK3196165 150mg or Tofacitinib 5mg BID from Day 1, received active intervention for 52 weeks.
Pre-assignment Details: Analysis of this study were reported for GSK3196165 90mg, GSK3196165 150mg, Tofacitinib 5 mg and all placebo arms are pooled to a single group to serve as reference for comparison of active treatment arms versus Placebo for primary efficacy endpoint analysis at Week 12.
Period: Overall Study
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX | Placebo + MTX and GSK3196165 90mg + MTX | Placebo + MTX and GSK3196165 150mg + MTX | Placebo + MTX and Tofacitinib 5mg + MTX
Started | 513 | 510 | 258 | 85 | 86 | 85
Safety Set (All randomized participants who received at least one dose of study treatment.) | 513 | 510 | 273 | 0 | 0 | 0
Safety Set-Placebo Switch (All participants randomized to a placebo switch treatment arm (i.e. Placebo to GSK3196165 90mg, Placebo to GSK3196165 150mg or Placebo to Tofacitinib 5mg) who received at least one dose of study treatment.) | 0 | 0 | 0 | 80 | 82 | 68
Completed | 431 | 436 | 221 | 69 | 73 | 75
Not Completed | 82 | 74 | 37 | 16 | 13 | 10
Not completed — Adverse Event | 13 | 29 | 11 | 2 | 2 | 2
Not completed — Lack of Efficacy | 7 | 6 | 0 | 3 | 1 | 1
Not completed — Lost to Follow-up | 2 | 4 | 2 | 1 | 2 | 0
Not completed — Protocol Violation | 4 | 2 | 1 | 1 | 0 | 0
Not completed — Physician Decision | 14 | 10 | 7 | 4 | 4 | 2
Not completed — Withdrawal by Subject | 38 | 21 | 15 | 5 | 3 | 4
Not completed — PROTOCOL-SPECIFIED WITHDRAWAL CRITERION MET | 4 | 0 | 1 | 0 | 1 | 1
Not completed — INVESTIGATOR SITE CLOSED | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX | Placebo + MTX and GSK3196165 90mg + MTX | Placebo + MTX and GSK3196165 150mg + MTX | Placebo + MTX and Tofacitinib 5mg + MTX | Total
Number analyzed (Participants) | 513 | 510 | 258 | 85 | 86 | 85 | 1537
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 53.7 (12.14) | 54.2 (10.77) | 54.3 (11.66) | 51.3 (13.12) | 52.7 (12.41) | 53.2 (10.24) | 53.8 (11.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 401 | 399 | 209 | 62 | 72 | 68 | 1211
  Male | 112 | 111 | 49 | 23 | 14 | 17 | 326
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  AMERICAN INDIAN OR ALASKA NATIVE | 11 | 11 | 9 | 2 | 3 | 2 | 38
  ASIAN | 48 | 39 | 29 | 5 | 7 | 4 | 132
  BLACK OR AFRICAN AMERICAN | 11 | 11 | 12 | 3 | 2 | 2 | 41
  MISSING | 1 | 0 | 0 | 1 | 1 | 1 | 4
  MULTIPLE | 10 | 15 | 7 | 2 | 2 | 1 | 37
  WHITE | 432 | 434 | 201 | 72 | 71 | 75 | 1285

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving 20 Percentage (%) Improvement in American College of Rheumatology Criteria (ACR20) at Week 12 Superiority Comparison With Placebo
Description: ACR20 is calculated as a 20% improvement from Baseline in Tender Joint Count 68 (TJC68) and Swollen Joint Count 66 (SJC66) and a 20% improvement in 3 of the following 5 measures: Patient's Global Assessment of Arthritis Disease Activity (PtGA) [visual analogue scale (VAS) with values from 0=best to 100=worst], Physician Global Assessment of Arthritis Disease Activity (PhGA) (VAS with values from 0=best to 100=worst), Patient Assessment of Arthritis Pain (VAS with values from 0=no pain and 100=most severe pain), Health Assessment Questionnaire-Disability Index (HAQ-DI) (ranges from 0 to 3 where 0 = least difficulty and 3 = extreme difficulty) and an acute-phase reactant [high sensitivity C-reactive Protein milligram per liter (mg/L) (hsCRP)]. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Week 12
Population: The analysis was performed on the Intent-to-Treat (ITT) set that inlcudes all randomized participants who received at least one dose of study treatment. This population was based on the treatment the participant was randomized to. Analysis was performed using multiple imputation method to handle missing data.
Measure: Number; unit: Percentage of participants
Groups:
- Pooled Placebo: Participants received Placebo weekly SC injection in combination with MTX until Week 12. The placebo arms are pooled into a single placebo arm.
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX | Pooled Placebo
Number analyzed (Participants) | 513 | 510 | 258 | 256
Percentage of participants | 54.7 | 50.9 | 63.6 | 42.7
Statistical Analysis 1: Comparison: GSK3196165 90mg + MTX vs Pooled Placebo; The null hypothesis is defined as there is no difference between the 90mg dose of GSK3196165 and placebo in the proportion of participants achieving ACR20 response at Week 12, versus the alternative hypothesis that the 90mg dose of GSK3196165 differs from placebo in the proportion of participants achieving ACR20 response at Week 12; Test type: Superiority; p = 0.0023, Regression, Logistic; OR and corresponding 95% CI for OR are generated from the logistic regression model adjusted for Baseline TJC68, Baseline SJC66 and Treatment Group; Odds Ratio (OR) = 1.62, .95% CI 2-sided [1.19 to 2.21]
Statistical Analysis 2: Comparison: GSK3196165 150mg + MTX vs Pooled Placebo; The null hypothesis is defined as there is no difference between the 150mg dose of GSK3196165 and placebo in the proportion of participants achieving ACR20 response at Week 12, versus the alternative hypothesis that the 150mg dose of GSK3196165 differs from placebo in the proportion of participants achieving ACR20 response at Week 12; Test type: Superiority; p = 0.0362, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.39, .95% CI 2-sided [1.02 to 1.89]
Statistical Analysis 3: Comparison: Tofacitinib 5mg + MTX vs Pooled Placebo; The null hypothesis is defined as there is no difference between the 05mg dose of Tofacitinib and placebo in the proportion of participants achieving ACR20 response at Week 12, versus the alternative hypothesis that the 05mg dose of Tofacitinib differs from placebo in the proportion of participants achieving ACR20 response at Week 12; Test type: Superiority; p < 0.0001, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.34, .95% CI 2-sided [1.62 to 3.37]
Statistical Analysis 4: Comparison: GSK3196165 90mg + MTX vs Tofacitinib 5mg + MTX; The null hypothesis is defined as there is no difference between the 90mg dose of GSK3196165 and 05mg dose of Tofacitinib in the proportion of participants achieving ACR20 response at Week 12, versus the alternative hypothesis that the 90mg dose of GSK3196165 differs from 05mg dose of Tofacitinib in the proportion of participants achieving ACR20 response at Week 12; Test type: Superiority; p = 0.0230, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.69, .95% CI 2-sided [0.50 to 0.95]
Statistical Analysis 5: Comparison: GSK3196165 150mg + MTX vs Tofacitinib 5mg + MTX; The null hypothesis is defined as there is no difference between the 150mg dose of GSK3196165 and 05mg dose of Tofacitinib in the proportion of participants achieving ACR20 response at Week 12, versus the alternative hypothesis that the 150mg dose of GSK3196165 differs from 05mg dose of Tofacitinib in the proportion of participants achieving ACR20 response at Week 12; Test type: Superiority; p = 0.0013, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.59, .95% CI 2-sided [0.43 to 0.82]

2. Secondary Outcome: Percentage of Participants Achieving Clinical Disease Activity Index (CDAI) Total Score Less Than or Equal to (<=)10 [CDAI Low Disease Activity (LDA)] at Week 12
Description: Clinical Disease Activity Index (CDAI) total score is a composite score consisting of the sum of Swollen Joint Count 28 (SJC28), Tender Joint Count 28 (TJC28), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst) and Physician Global Assessment of Arthritis Disease Activity (PhGA) (visual analogue scale with values from 0=best to 100=worst). PtGA and PhGA are transformed to a 0-10 scale before computing the CDAI total score. CDAI total score ranges from 0 to 76 with higher values representing higher disease activity. Low disease activity (LDA) is achieved when CDAI total score <=10. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Week 12
Population: The analysis was performed on the ITT set that inlcudes all randomized participants who received at least one dose of study treatment. This population was based on the treatment the participant was randomized to. Analysis was performed using multiple imputation method to handle missing data.
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX | Pooled Placebo
Number analyzed (Participants) | 513 | 510 | 258 | 256
Percentage of participants | 20.9 | 19.8 | 32.5 | 13.9

3. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) at Week 12
Description: Health Assessment Questionnaire-Disability Index (HAQ-DI) is a 20-question instrument that assesses degree of difficulty of a participant in accomplishing tasks in eight functional areas: dressing and grooming, arising, eating, walking, hygiene, reach, grip and common daily activities. Overall HAQ-DI score was computed as sum of the domain scores divided by the number of domains answered. The total possible score ranges from 0 to 3 where 0=least difficulty and 3=extreme difficulty. Higher overall score indicates greater disability. A negative change from baseline indicates an improvement. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX | Pooled Placebo
Number analyzed (Participants) | 513 | 510 | 258 | 256
Scores on a scale | -0.46 (0.025) | -0.38 (0.024) | -0.5 (0.034) | -0.27 (0.034)

4. Secondary Outcome: Percentage of Participants Achieving 20% Improvement in ACR20 at Week 24 (Non-Inferiority Versus Tofacitinib)
Description: ACR20 is calculated as a 20% improvement from Baseline in Tender Joint Count 68 (TJC68) and Swollen Joint Count 66 (SJC66) and a 20% improvement in 3 of the following 5 measures: Patient's Global Assessment of Arthritis Disease Activity (PtGA) [visual analogue scale (VAS) with values from 0=best to 100=worst], Physician Global Assessment of Arthritis Disease Activity (PhGA) (VAS with values from 0=best to 100=worst), Patient Assessment of Arthritis Pain (VAS with values from 0=no pain and 100=most severe pain), Health Assessment Questionnaire-Disability Index (HAQ-DI) (ranges from 0 to 3 where 0 = least difficulty and 3 = extreme difficulty) and an acute-phase reactant [high sensitivity C-reactive Protein milligram per liter (mg/L) (hsCRP)].
Time Frame: Week 24
Population: The analysis was performed on the ITT set that includes all randomized participants who received at least one dose of study treatment. This population was based on the treatment the subject was randomized to. Analysis was performed using multiple imputation method to handle missing data.
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX
Number analyzed (Participants) | 513 | 510 | 258
Percentage of participants | 63.9 | 61.3 | 74.4
Statistical Analysis 1: Comparison: GSK3196165 90mg + MTX vs Tofacitinib 5mg + MTX; Test type: Non-Inferiority — Non-inferiority over tofacitinib on ACR20 was concluded if the lower limit of the multiplicity corrected 97.5 % Confidence Interval (CI) in the difference in proportions (GSK3196165 minus tofacitinib) was greater than -12%; Regression, Logistic; Difference in proportion and 97.5% CI are generated from logistic regression model adjusted for Baseline TJC68, Baseline SJC66 and Treatment Group; Mean Difference (Final Values) = -10.4, .975% CI 2-sided [-18.6 to -2.3]
Statistical Analysis 2: Comparison: GSK3196165 150mg + MTX vs Tofacitinib 5mg + MTX; Test type: Non-Inferiority — Non-inferiority over tofacitinib on ACR20 was concluded if the lower limit of the multiplicity corrected 97.5% CI in the difference in proportions (GSK3196165 minus tofacitinib) was greater than -12%; Regression, Logistic; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -13.0, .975% CI 2-sided [-21.2 to -4.8]

5. Secondary Outcome: Percentage of Participants Achieving 50%/70% Improvement in American College of Rheumatology Criteria (ACR50/70) at Week 24 and ACR 20/50/70 at and Week 52 for Treatment Arms Who Started Study Intervention From Day 1
Description: ACR20/50/70 is calculated as a 20%/50%/70% improvement from Baseline in Tender Joint Count 68 (TJC68) and Swollen Joint Count 66 (SJC66) and a 20%/50%/70% improvement in 3 of the following 5 measures: Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale (VAS) with values from 0=best to 100=worst), Physician Global Assessment of Arthritis Disease Activity (PhGA) [VAS with values from 0=best to 100=worst], Patient Assessment of Arthritis Pain (VAS with values from 0=no pain and 100=most severe pain), Health Assessment Questionnaire-Disability Index (HAQ- DI) (ranges from 0 to 3 where 0 = least difficulty and 3 = extreme difficulty) and an acute-phase reactant [high sensitivity C-reactive Protein mg/L (hsCRP)].
Time Frame: Week 24 and Week 52
Population: The analysis was performed on all randomized participants who received study intervention from Day 01 to Week 52. Analysis was performed using multiple imputation method to handle missing data.
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX
Number analyzed (Participants) | 513 | 510 | 258
Percentage of participants
  ACR20, Week 52 | 63.9 | 61.1 | 75.8
  ACR50, Week 24 | 31.4 | 29.1 | 46.7
  ACR50, Week 52 | 35.0 | 34.2 | 48.4
  ACR70, Week 24 | 12.5 | 10.1 | 25.1
  ACR70, Week 52 | 16.7 | 14.4 | 26.9

6. Secondary Outcome: Percentage of Participants Achieving ACR20/50/70 at Week 24 and Week 52 for Placebo Switched Arms
Description: as for outcome 5
Time Frame: Week 24 and Week 52
Population: The analysis was performed on all randomized participants who switched from placebo to study intervention at Week 12. Analysis was performed using multiple imputation method to handle missing data.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + MTX and GSK3196165 90mg + MTX | Placebo + MTX and GSK3196165 150mg + MTX | Placebo + MTX and Tofacitinib 5mg + MTX
Number analyzed (Participants) | 85 | 86 | 85
Percentage of participants
  ACR20, Week 24 | 56.7 | 71.2 | 69.9
  ACR20, Week 52 | 70.5 | 67.8 | 84.6
  ACR50, Week 24 | 37.0 | 35.0 | 40.7
  ACR50, Week 52 | 28.6 | 42.5 | 50.7
  ACR70, Week 24 | 7.9 | 15.0 | 19.6
  ACR70, Week 52 | 10.3 | 20.2 | 25.8

7. Secondary Outcome: Percentage of Participants Achieving CDAI Total Score <=10 (CDAI LDA) at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1
Description: Clinical Disease Activity Index (CDAI) total score is a composite score consisting of the sum of Swollen Joint Count 28 (SJC28), Tender Joint Count 28 (TJC28), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst) and Physician Global Assessment of Arthritis Disease Activity (PhGA) (visual analogue scale with values from 0=best to 100=worst). PtGA and PhGA are transformed to a 0-10 scale before computing the CDAI total score. CDAI total score ranges from 0 to 76 with higher values representing higher disease activity. Low disease activity (LDA) is achieved when CDAI total score <=10.
Time Frame: Week 24 and Week 52
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX
Number analyzed (Participants) | 513 | 510 | 258
Percentage of participants
  Week 24 | 29.9 | 29.8 | 45.9
  Week 52 | 35.5 | 37.1 | 51.7

8. Secondary Outcome: Percentage of Participants Achieving CDAI Total Score <=10 (CDAI LDA) at Week 24 and Week 52 for Placebo Switched Arms
Description: as for outcome 7
Time Frame: Week 24 and Week 52
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + MTX and GSK3196165 90mg + MTX | Placebo + MTX and GSK3196165 150mg + MTX | Placebo + MTX and Tofacitinib 5mg + MTX
Number analyzed (Participants) | 85 | 86 | 85
Percentage of participants
  Week 24 | 32.9 | 37.4 | 45.8
  Week 52 | 38.5 | 44 | 52.4

9. Secondary Outcome: Percentage of Participants Achieving CDAI Total Score <=2.8 (CDAI Remission) at Week 12
Description: Clinical Disease Activity Index (CDAI) total score is a composite score consisting of the sum of Swollen Joint Count 28 (SJC28), Tender Joint Count 28 (TJC28), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst) and Physician Global Assessment of Arthritis Disease Activity (PhGA) (visual analogue scale with values from 0=best to 100=worst). PtGA and PhGA are transformed to a 0-10 scale before computing the CDAI total score. CDAI total score ranges from 0 to 76 with higher values representing higher disease activity. CDAI remission is achieved when CDAI total score <=2.8. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX | Pooled Placebo
Number analyzed (Participants) | 513 | 510 | 258 | 256
Percentage of participants | 3.8 | 2.4 | 5.8 | 1.0

10. Secondary Outcome: Percentage of Participants Achieving CDAI Total Score <=2.8 (CDAI Remission) at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1
Description: Clinical Disease Activity Index (CDAI) total score is a composite score consisting of the sum of Swollen Joint Count 28 (SJC28), Tender Joint Count 28 (TJC28), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst) and Physician Global Assessment of Arthritis Disease Activity (PhGA) (visual analogue scale with values from 0=best to 100=worst). PtGA and PhGA are transformed to a 0-10 scale before computing the CDAI total score. CDAI total score ranges from 0 to 76 with higher values representing higher disease activity. CDAI remission is achieved when CDAI total score <=2.8.
Time Frame: Week 24 and Week 52
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX
Number analyzed (Participants) | 513 | 510 | 258
Percentage of participants
  Week 24 | 6.1 | 5.2 | 12.1
  Week 52 | 9.4 | 4.4 | 15.1

11. Secondary Outcome: Percentage of Participants Achieving CDAI Total Score <=2.8 (CDAI Remission) at Week 24 and Week 52 for Placebo Switched Arms
Description: as for outcome 10
Time Frame: Week 24 and Week 52
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + MTX and GSK3196165 90mg + MTX | Placebo + MTX and GSK3196165 150mg + MTX | Placebo + MTX and Tofacitinib 5mg + MTX
Number analyzed (Participants) | 85 | 86 | 85
Percentage of participants
  Week 24 | 4.4 | 8.4 | 6.4
  Week 52 | 4.6 | 9.6 | 11.1

12. Secondary Outcome: Percentage of Participants Achieving 50%/70% Improvement in American College of Rheumatology Criteria (ACR50/70) at Week 12
Description: ACR50/70 is calculated as a 50%/70% improvement from Baseline in Tender Joint Count 68 (TJC68) and Swollen Joint Count 66 (SJC66) and a 50%/70% improvement in 3 of the following 5 measures: Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale (VAS) with values from 0=best to 100=worst), Physician Global Assessment of Arthritis Disease Activity (PhGA) [VAS with values from 0=best to 100=worst), Patient Assessment of Arthritis Pain (VAS with values from 0=no pain and 100=most severe pain), Health Assessment Questionnaire-Disability Index (HAQ-DI) (ranges from 0 to 3 where 0 = least difficulty and 3 = extreme difficulty) and an acute-phase reactant (high sensitivity C-reactive Protein mg/L (hsCRP)]. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX | Pooled Placebo
Number analyzed (Participants) | 513 | 510 | 258 | 256
Percentage of participants
  ACR50, Week 12 | 23.3 | 20.0 | 34.1 | 12.2
  ACR70, Week 12 | 8.5 | 6.1 | 13.9 | 3.5

13. Secondary Outcome: Percentage of Participants Achieving Disease Activity Score Using 28 Joint Count and C-Reactive Protein (DAS28-CRP) <=3.2 (DAS28-CRP LDA) at Week 12
Description: The DAS28-CRP is a measure of RA disease activity calculated using Tender Joint Count 28 (TJC28), Swollen Joint Count 28 (SJC28), C-reactive protein (CRP) (in mg/L), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst). DAS28- CRP scores range from 1.0 to 9.4, where lower scores indicate less disease activity. Low disease activity (LDA) is achieved when DAS28-CRP greater than or equal to (<=)3.2. A negative change from baseline in DAS28-CRP indicates an improvement. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX | Pooled Placebo
Number analyzed (Participants) | 513 | 510 | 258 | 256
Percentage of participants | 20.2 | 19.4 | 33.5 | 11.3

14. Secondary Outcome: Percentage of Participants Achieving DAS28 Erythrocyte Sedimentation Rate (ESR) <=3.2 (DAS28-ESR LDA) at Week 12
Description: The DAS28-ESR is a measure of RA disease activity calculated using Tender Joint Count 28 (TJC28), Swollen Joint Count 28 (SJC28), Erythrocyte sedimentation rate (ESR) (in millimeter [mm]/hour[hr]), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst). DAS28-ESR scores range from 1.0 to 9.4, where lower scores indicate less disease activity. Low disease activity (LDA) is achieved when DAS28-ESR<=3.2. A negative change from baseline in DAS28-ESR indicates an improvement. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX | Pooled Placebo
Number analyzed (Participants) | 513 | 510 | 258 | 256
Percentage of participants | 13.6 | 12.2 | 19.7 | 8.2

15. Secondary Outcome: Percentage of Participants Achieving DAS28-CRP <=3.2 (DAS28-CRP LDA) at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1
Description: The DAS28-CRP is a measure of RA disease activity calculated using Tender Joint Count 28 (TJC28), Swollen Joint Count 28 (SJC28), C-reactive protein (CRP) (in mg/L), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst). DAS28-CRP scores range from 1.0 to 9.4, where lower scores indicate less disease activity. Low disease activity (LDA) is achieved when DAS28-CRP<=3.2. A negative change from baseline in DAS28-CRP indicates an improvement.
Time Frame: Week 24 and Week 52
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX
Number analyzed (Participants) | 513 | 510 | 258
Percentage of participants
  Week 24 | 26.8 | 29.0 | 47.4
  Week 52 | 32.8 | 31.3 | 49.8

16. Secondary Outcome: Percentage of Participants Achieving DAS28-ESR <=3.2 (DAS28-ESR LDA) at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1
Description: The DAS28-ESR is a measure of RA disease activity calculated using Tender Joint Count 28 (TJC28), Swollen Joint Count 28 (SJC28), Erythrocyte sedimentation rate (ESR) (in millimeter [mm]/hour[hr]), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst). DAS28-ESR scores range from 1.0 to 9.4, where lower scores indicate less disease activity. Low disease activity (LDA) is achieved when DAS28-ESR<=3.2. A negative change from baseline in DAS28-ESR indicates an improvement.
Time Frame: Week 24 and Week 52
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX
Number analyzed (Participants) | 513 | 510 | 258
Percentage of participants
  Week 24 | 17.2 | 18.3 | 28.3
  Week 52 | 23.3 | 18.7 | 34.1

17. Secondary Outcome: Percentage of Participants Achieving DAS28-CRP <=3.2 (DAS28-CRP LDA) at Week 24 and Week 52 for Placebo Switched Arms
Description: as for outcome 15
Time Frame: Week 24 and Week 52
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + MTX and GSK3196165 90mg + MTX | Placebo + MTX and GSK3196165 150mg + MTX | Placebo + MTX and Tofacitinib 5mg + MTX
Number analyzed (Participants) | 85 | 86 | 85
Percentage of participants
  Week 24 | 26.3 | 31.0 | 44.9
  Week 52 | 34.2 | 34.9 | 50.2

18. Secondary Outcome: Percentage of Participants Achieving DAS28-ESR <=3.2 (DAS28-ESR LDA) at Week 24 and Week 52 for Placebo Switched Arms
Description: as for outcome 16
Time Frame: Week 24 and Week 52
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + MTX and GSK3196165 90mg + MTX | Placebo + MTX and GSK3196165 150mg + MTX | Placebo + MTX and Tofacitinib 5mg + MTX
Number analyzed (Participants) | 85 | 86 | 85
Percentage of participants
  Week 24 | 20.7 | 22.7 | 30.4
  Week 52 | 22.9 | 21.8 | 30.3

19. Secondary Outcome: Percentage of Participants Achieving DAS28-CRP <2.6 (DAS28-CRP Remission) at Week 12
Description: The DAS28-CRP is a measure of RA disease activity calculated using Tender Joint Count 28 (TJC28), Swollen Joint Count 28 (SJC28), C-reactive protein (CRP) (in mg/L), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst). DAS28-CRP scores range from 1.0 to 9.4, where lower scores indicate less disease activity. Remission is achieved when DAS28-CRP less than (<)2.6. A negative change from baseline in DAS28-CRP indicates an improvement. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX | Pooled Placebo
Number analyzed (Participants) | 513 | 510 | 258 | 256
Percentage of participants | 10.3 | 8.4 | 17.1 | 5.2

20. Secondary Outcome: Percentage of Participants Achieving DAS28 ESR <2.6 (DAS28-ESR Remission) at Week 12
Description: The DAS28-ESR is a measure of RA disease activity calculated using Tender Joint Count 28 (TJC28), Swollen Joint Count 28 (SJC28), Erythrocyte sedimentation rate (ESR) (in mm/hr), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst). DAS28-ESR scores range from 1.0 to 9.4, where lower scores indicate less disease activity. Remission is achieved when DAS28-ESR <2.6. A negative change from baseline in DAS28-ESR indicates an improvement. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX | Pooled Placebo
Number analyzed (Participants) | 513 | 510 | 258 | 256
Percentage of participants | 6.0 | 5.3 | 11.5 | 5.2

21. Secondary Outcome: Percentage of Participants Achieving DAS28-CRP <2.6 (DAS28-CRP Remission) at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1
Description: The DAS28-CRP is a measure of RA disease activity calculated using Tender Joint Count 28 (TJC28), Swollen Joint Count 28 (SJC28), C-reactive protein (CRP) (in mg/L), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst). DAS28-CRP scores range from 1.0 to 9.4, where lower scores indicate less disease activity. Remission is achieved when DAS28-CRP <2.6. A negative change from baseline in DAS28-CRP indicates an improvement.
Time Frame: Week 24 and Week 52
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX
Number analyzed (Participants) | 513 | 510 | 258
Percentage of participants
  Week 24 | 14.5 | 14.1 | 26.3
  Week 52 | 19.3 | 15.3 | 34.0

22. Secondary Outcome: Percentage of Participants Achieving DAS28 ESR <2.6 (DAS28-ESR Remission) at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1
Description: The DAS28-ESR is a measure of RA disease activity calculated using Tender Joint Count 28 (TJC28), Swollen Joint Count 28 (SJC28), Erythrocyte sedimentation rate (ESR) (in mm/hr), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst). DAS28-ESR scores range from 1.0 to 9.4, where lower scores indicate less disease activity. Remission is achieved when DAS28-ESR <2.6. A negative change from baseline in DAS28-ESR indicates an improvement.
Time Frame: Week 24 and Week 52
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX
Number analyzed (Participants) | 513 | 510 | 258
Percentage of participants
  Week 24 | 8.6 | 7.8 | 13.7
  Week 52 | 14.1 | 8.8 | 18.7

23. Secondary Outcome: Percentage of Participants Achieving DAS28-CRP <2.6 (DAS28-CRP Remission) at Week 24 and Week 52 for Placebo Switched Arms
Description: as for outcome 21
Time Frame: Week 24 and Week 52
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + MTX and GSK3196165 90mg + MTX | Placebo + MTX and GSK3196165 150mg + MTX | Placebo + MTX and Tofacitinib 5mg + MTX
Number analyzed (Participants) | 85 | 86 | 85
Percentage of participants
  Week 24 | 14.7 | 20.2 | 28.2
  Week 52 | 18.2 | 18.7 | 31.2

24. Secondary Outcome: Percentage of Participants Achieving DAS28 ESR <2.6 (DAS28-ESR Remission) at Week 24 and Week 52 for Placebo Switched Arms
Description: as for outcome 22
Time Frame: Week 24 and Week 52
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + MTX and GSK3196165 90mg + MTX | Placebo + MTX and GSK3196165 150mg + MTX | Placebo + MTX and Tofacitinib 5mg + MTX
Number analyzed (Participants) | 85 | 86 | 85
Percentage of participants
  Week 24 | 10.8 | 14.8 | 12
  Week 52 | 11.0 | 11.8 | 15.5

25. Secondary Outcome: Percentage of Participants Achieving a Good/Moderate (European League Against Rheumatism) EULAR Response at Week 12
Description: DAS28-CRP and DAS28-ESR scores were categorized using EULAR response criteria. Response at given time point was defined based on the combination of current DAS28 score and improvement in the current DAS28 score relative to Baseline. The definition of no response, moderate response and good response was as; DAS28 <=3.2 and DAS28 decrease from Baseline (>1.2:good response), (>0.6 to <=1.2:moderate response) and (<=0.6:no response); DAS28 >3.2 to <=5.1 and DAS28 decrease from Baseline (>1.2:moderate response), (>0.6 to <=1.2:moderate response) and (<=0.6:no response) and DAS28 >5.1 and DAS28 decrease from Baseline (>1.2:moderate response), (>0.6 to <=1.2:no response) and (<=0.6:no response). If the post-Baseline DAS28-CRP score was missing, then the corresponding EULAR category was set to missing. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX | Pooled Placebo
Number analyzed (Participants) | 513 | 510 | 258 | 256
Percentage of participants | 73.1 | 69.3 | 83.0 | 54.5

26. Secondary Outcome: Percentage of Participants Achieving a Good/Moderate EULAR Response at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1
Description: DAS28-CRP and DAS28-ESR scores were categorized using EULAR response criteria. Response at a given time point was defined based on the combination of current DAS28 score and the improvement in the current DAS28 score relative to Baseline. The definition of no response, moderate response and good response was as; if current DAS28 <=3.2 and DAS28 decrease from Baseline (>1.2: good response), (>0.6 to <=1.2: moderate response) and (<=0.6: no response); if current DAS28 >3.2 to <=5.1 and DAS28 decrease from Baseline value (>1.2: moderate response), (>0.6 to <=1.2: moderate response) and (<=0.6: no response) and if current DAS28 >5.1 and DAS28 decrease from Baseline value (>1.2: moderate response), (>0.6 to <=1.2: no response) and (<=0.6: no response). If the post-Baseline DAS28-CRP score was missing, then the corresponding EULAR category was set to missing.
Time Frame: Week 24 and Week 52
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX
Number analyzed (Participants) | 513 | 510 | 258
Percentage of participants
  Week 24 | 78.4 | 74.9 | 89.8
  Week 52 | 79.1 | 78.6 | 89.0

27. Secondary Outcome: Percentage of Participants Achieving a Good/Moderate EULAR Response at Week 24 and Week 52 for Placebo Switched Arms
Description: as for outcome 26
Time Frame: Week 24 and Week 52
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + MTX and GSK3196165 90mg + MTX | Placebo + MTX and GSK3196165 150mg + MTX | Placebo + MTX and Tofacitinib 5mg + MTX
Number analyzed (Participants) | 85 | 86 | 85
Percentage of participants
  Week 24 | 76.3 | 82.4 | 88.9
  Week 52 | 87.1 | 79.1 | 92.5

28. Secondary Outcome: Number of Participants Achieving ACR/EULAR Remission at Week 12
Description: Boolean-based ACR/EULAR remission is achieved if all of the following requirements are met at the same timepoint: Tender Joint Count 68 (TJC68) <= 1, Swollen Joint Count 66 (SJC66) <= 1, high sensitivity C-reactive Protein (hsCRP) <= 1mg/dl and patient's global assessment of disease activity (PtGA) <= 10. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Week 12
Population: The analysis was performed on the ITT set that inlcudes all randomized participants who received at least one dose of study treatment. This population was based on the treatment the participant was randomized to. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX | Pooled Placebo
Number analyzed (Participants) | 475 | 477 | 228 | 235
Participants | 11 | 9 | 11 | 2

29. Secondary Outcome: Number of Participants Achieving ACR/EULAR Remission at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1
Description: Boolean-based ACR/EULAR remission is achieved if all of the following requirements are met at the same timepoint: Tender Joint Count 68 (TJC68) <= 1, Swollen Joint Count 66 (SJC66) <= 1, high sensitivity C-reactive Protein (hsCRP) <= 1mg/dl and patient's global assessment of disease activity (PtGA) <= 10.
Time Frame: Week 24 and Week 52
Population: The analysis was performed on all randomized participants who received study intervention from Day 01 to Week 52. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX
Number analyzed (Participants) | 453 | 467 | 227
Participants
  Week 24 | 16 | 13 | 14
  Week 52: number analyzed (Participants) | 416 | 420 | 209
  Week 52 | 24 | 13 | 18

30. Secondary Outcome: Number of Participants Achieving ACR/EULAR Remission at Week 24 and Week 52 for Placebo Switched Arms
Description: as for outcome 29
Time Frame: Week 24 and Week 52
Population: The analysis was performed on all randomized participants who switched from placebo to study intervention at Week 12. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + MTX and GSK3196165 90mg + MTX | Placebo + MTX and GSK3196165 150mg + MTX | Placebo + MTX and Tofacitinib 5mg + MTX
Number analyzed (Participants) | 76 | 80 | 78
Participants
  Week 24 | 2 | 4 | 3
  Week 52: number analyzed (Participants) | 67 | 71 | 74
  Week 52 | 3 | 3 | 8

31. Secondary Outcome: Percentage of Participants Achieving no Radiographic Progression (Van Der Heijde Modified Total Sharp Scores (mTSS <= 0.5) at Week 12
Description: Van der Heijde mTSS is utilized for scoring radiographs of hands and feet in rheumatoid arthritis. This method includes 16 areas of erosions, and 15 areas for joint space narrowing (JSN) in each hand, and 6 areas for erosions and 6 areas JSN in each foot. The total mTSS score is the sum of erosion (maximum of 280) and JSN (maximum of 168) scores. The score ranges from 0 to 448 for mTSS with higher values representing higher disease activity. No radiographic progression is defined as a change from Baseline in van der Heijde mTSS score of <=0.5. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Week 12
Population: The analysis was performed on the ITT set that inlcudes all randomized participants who received at least one dose of study treatment. This population was based on the treatment the subject was randomized to. Analysis was performed using multiple imputation method to handle missing data.
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX | Pooled Placebo
Number analyzed (Participants) | 513 | 510 | 258 | 256
Percentage of participants | 83.8 | 82.6 | 88.9 | 76.7

32. Secondary Outcome: Percentage of Participants Achieving no Radiographic Progression (mTSS <= 0.5) at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1
Description: Van der Heijde mTSS is utilized for scoring radiographs of hands and feet in rheumatoid arthritis. This method includes 16 areas of erosions, and 15 areas for joint space narrowing (JSN) in each hand, and 6 areas for erosions and 6 areas JSN in each foot. The total mTSS score is the sum of erosion (maximum of 280) and JSN (maximum of 168) scores. The score ranges from 0 to 448 for mTSS with higher values representing higher disease activity. No radiographic progression is defined as a change from Baseline in van der Heijde mTSS score of <=0.5.
Time Frame: Week 24 and Week 52
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX
Number analyzed (Participants) | 513 | 510 | 258
Percentage of participants
  mTSS <= 0.5, Week 24 | 79.5 | 79.6 | 84.6
  mTSS <= 0.5, Week 52 | 71.8 | 72.8 | 79.7

33. Secondary Outcome: Percentage of Participants Achieving no Radiographic Progression (mTSS <= 0.5) at Week 24 and Week 52 for Placebo Switched Arms
Description: as for outcome 32
Time Frame: Week 24 and Week 52
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + MTX and GSK3196165 90mg + MTX | Placebo + MTX and GSK3196165 150mg + MTX | Placebo + MTX and Tofacitinib 5mg + MTX
Number analyzed (Participants) | 85 | 86 | 85
Percentage of participants
  mTSS <= 0.5, Week 24 | 78.6 | 74.6 | 77.7
  mTSS <= 0.5, Week 52 | 76.0 | 68.3 | 69.5

34. Secondary Outcome: Change From Baseline in CDAI Total Score at Week 12
Description: Clinical Disease Activity Index (CDAI) total score is a composite score consisting of sum of Swollen Joint Count 28 (SJC28), Tender Joint Count 28 (TJC28), Patient's Global Assessment of Arthritis Disease Activity (PtGA) and Physician Global Assessment of Arthritis Disease Activity (PhGA) (PtGA and PhGA VAS with values from 0=best to 100=worst). PtGA and PhGA are transformed to a 0-10 scale before computing the CDAI total score. CDAI total score ranges from 0 to 76 with higher values representing higher disease activity. Low disease activity (LDA) is achieved when CDAI total score <=10. Baseline was defined as latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting post dose visit value from Baseline value. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX | Pooled Placebo
Number analyzed (Participants) | 513 | 510 | 258 | 256
Scores on a scale | -17.85 (0.574) | -17.15 (0.563) | -21.39 (0.801) | -13.01 (0.798)

35. Secondary Outcome: Change From Baseline in CDAI Total Score at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1
Description: CDAI total score is a composite score consisting of the sum of Swollen Joint Count 28 (SJC28), Tender Joint Count 28 (TJC28), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst) and Physician Global Assessment of Arthritis Disease Activity (PhGA) (visual analogue scale with values from 0=best to 100=worst). PtGA and PhGA are transformed to a 0-10 scale before computing the CDAI total score. CDAI total score ranges from 0 to 76 with higher values representing higher disease activity. Low disease activity (LDA) is achieved when CDAI total score <=10. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX
Number analyzed (Participants) | 513 | 510 | 258
Scores on a scale
  Week 24 | -20.63 (0.561) | -19.88 (0.551) | -24.5 (0.781)
  Week 52 | -21.79 (0.558) | -21.81 (0.549) | -25.55 (0.77)

36. Secondary Outcome: Change From Baseline in CDAI Total Score at Week 24 and Week 52 for Placebo Switched Arms
Description: CDAI total score is a composite score consisting of the sum of Swollen Joint Count 28 (SJC28), Tender Joint Count 28 (TJC28), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst) and Physician Global Assessment of Arthritis Disease Activity (PhGA) (visual analogue scale with values from 0=best to 100=worst). PtGA and PhGA are transformed to a 0-10 scale before computing the CDAI total score. CDAI total score ranges from 0 to 76 with higher values representing higher disease activity. Low disease activity (LDA) is achieved when CDAI total score <=10. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For efficacy assessments baseline is interpreted as Day 1.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo + MTX and GSK3196165 90mg + MTX | Placebo + MTX and GSK3196165 150mg + MTX | Placebo + MTX and Tofacitinib 5mg + MTX
Number analyzed (Participants) | 85 | 86 | 85
Scores on a scale
  Week 24 | -21.41 (1.359) | -22.93 (1.31) | -24.5 (1.307)
  Week 52 | -23.49 (1.365) | -22.91 (1.291) | -25.83 (1.28)

37. Secondary Outcome: Change From Baseline in DAS28-CRP/DAS28-ESR at Week 12
Description: DAS28-CRP and DAS28-ESR are measure of RA disease activity calculated using Swollen Joint Count 28 (SJC28), Tender Joint Count 28 (TJC28), high sensitivity C-reactive Protein (hsCRP in mg/L)/Erythrocyte sedimentation rate (ESR) [ESR in millimeter/hour (mm/hr)] and patient's global assessment of disease activity (PtGA) transformed to a 0-10 scale. Total score range from 0-9.4, with higher scores indicating more disease activity. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX | Pooled Placebo
Number analyzed (Participants) | 513 | 510 | 258 | 256
Scores on a scale
  DAS28-CRP | -1.49 (0.054) | -1.44 (0.053) | -1.96 (0.076) | -1.01 (0.075)
  DAS28-ESR | -1.53 (0.057) | -1.48 (0.056) | -1.97 (0.079) | -1.07 (0.079)

38. Secondary Outcome: Change From Baseline in DAS28-CRP/DAS28-ESR at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1
Description: DAS28-CRP and DAS28-ESR are measure of RA disease activity calculated using Swollen Joint Count 28 (SJC28), Tender Joint Count 28 (TJC28), high sensitivity C-reactive Protein (hsCRP in mg/L)/Erythrocyte sedimentation rate (ESR) [ESR in millimeter/hour (mm/hr)] and patient's global assessment of disease activity (PtGA) transformed to a 0-10 scale. Total score approximate range 0-9.4, with higher scores indicating more disease activity. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX
Number analyzed (Participants) | 513 | 510 | 258
Scores on a scale
  DAS28-CRP, Week 24 | -1.74 (0.056) | -1.67 (0.055) | -2.31 (0.078)
  DAS28-CRP, Week 52 | -1.85 (0.06) | -1.82 (0.059) | -2.39 (0.083)
  DAS28-ESR, Week 24 | -1.79 (0.059) | -1.74 (0.057) | -2.3 (0.082)
  DAS28-ESR, Week 52 | -1.92 (0.063) | -1.84 (0.062) | -2.36 (0.087)

39. Secondary Outcome: Change From Baseline in DAS28-CRP/DAS28-ESR at Week 24 and Week 52 for Placebo Switched Arms
Description: DAS28-CRP and DAS28-ESR are measure of RA disease activity calculated using Swollen Joint Count 28 (SJC28), Tender Joint Count 28 (TJC28), high sensitivity C-reactive Protein (hsCRP in mg/L)/Erythrocyte sedimentation rate (ESR) [ESR in millimeter/hour (mm/hr)] and patient's global assessment of disease activity (PtGA) transformed to a 0-10 scale. Total score approximate range 0-9.4, with higher scores indicating more disease activity. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For efficacy assessments baseline is interpreted as Day 1.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo + MTX and GSK3196165 90mg + MTX | Placebo + MTX and GSK3196165 150mg + MTX | Placebo + MTX and Tofacitinib 5mg + MTX
Number analyzed (Participants) | 85 | 86 | 85
Scores on a scale
  DAS28-CRP, Week 24 | -1.77 (0.136) | -1.95 (0.131) | -2.29 (0.131)
  DAS28-CRP, Week 52 | -1.92 (0.146) | -1.96 (0.139) | -2.37 (0.137)
  DAS28-ESR, Week 24 | -1.84 (0.143) | -2.05 (0.137) | -2.23 (0.137)
  DAS28-ESR, Week 52 | -2.06 (0.151) | -2.06 (0.145) | -2.43 (0.145)

40. Secondary Outcome: Change From Baseline in Van Der Heijde mTSS at Week 12
Description: Van der Heijde mTSS is utilized for scoring radiographs of hands and feet in rheumatoid arthritis. This method includes 16 areas of erosions, and 15 areas for joint space narrowing (JSN) in each hand, and 6 areas for erosions and 6 areas JSN in each foot. The total mTSS score is the sum of erosion (maximum of 280) and JSN (maximum of 168) scores. The score range from 0 to 448 for mTSS with higher values representing higher disease activity. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 1) and Week 12
Population: The analysis was performed on the ITT set that inlcude all randomized participants who received at least one dose of study treatment. This population was based on the treatment the participant was randomized to. Analysis was performed using multiple imputation method to handle missing data.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX | Pooled Placebo
Number analyzed (Participants) | 513 | 510 | 258 | 256
Scores on a scale | 0.15 (0.075) | 0.19 (0.073) | 0.13 (0.104) | 0.55 (0.103)

41. Secondary Outcome: Change From Baseline in Van Der Heijde mTSS at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1
Description: Van der Heijde mTSS is utilized for scoring radiographs of hands and feet in rheumatoid arthritis. This method includes 16 areas of erosions, and 15 areas for joint space narrowing (JSN) in each hand, and 6 areas for erosions and 6 areas JSN in each foot. The total mTSS score is the sum of erosion (maximum of 280) and JSN (maximum of 168) scores. The score range from 0 to 448 for mTSS with higher values representing higher disease activity. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX
Number analyzed (Participants) | 513 | 510 | 258
Scores on a scale
  Week 24 | 0.25 (0.08) | 0.38 (0.078) | 0.2 (0.112)
  Week 52 | 0.61 (0.117) | 0.63 (0.114) | 0.35 (0.158)

42. Secondary Outcome: Change From Baseline in Van Der Heijde mTSS at Week 24 and Week 52 for Placebo Switched Arms
Description: Van der Heijde mTSS is utilized for scoring radiographs of hands and feet in rheumatoid arthritis. This method includes 16 areas of erosions, and 15 areas for joint space narrowing (JSN) in each hand, and 6 areas for erosions and 6 areas JSN in each foot. The total mTSS score is the sum of erosion (maximum of 280) and JSN (maximum of 168) scores. The score range from 0 to 448 for mTSS with higher values representing higher disease activity. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For efficacy assessments baseline is interpreted as Day 1.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo + MTX and GSK3196165 90mg + MTX | Placebo + MTX and GSK3196165 150mg + MTX | Placebo + MTX and Tofacitinib 5mg + MTX
Number analyzed (Participants) | 85 | 86 | 85
Scores on a scale
  Week 24 | 0.71 (0.215) | 0.77 (0.208) | 0.67 (0.208)
  Week 52 | 0.9 (0.309) | 1.24 (0.306) | 1.06 (0.297)

43. Secondary Outcome: Change From Baseline in HAQ-DI at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1
Description: HAQ-DI is a 20-question instrument that assesses the degree of difficulty of a participant in accomplishing tasks in eight functional areas: dressing and grooming, arising, eating, walking, hygiene, reach, grip and common daily activities. Overall HAQ-DI score was computed as sum of the domain scores divided by the number of domains answered. The total possible score ranges from 0 to 3 where 0 = least difficulty and 3 = extreme difficulty. Higher overall score indicates greater disability. A negative change from baseline indicates an improvement. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX
Number analyzed (Participants) | 513 | 510 | 258
Scores on a scale
  Week 24 | -0.51 (0.027) | -0.41 (0.026) | -0.56 (0.037)
  Week 52 | -0.54 (0.028) | -0.46 (0.028) | -0.58 (0.039)

44. Secondary Outcome: Change From Baseline in HAQ-DI at Week 24 and Week 52 for Placebo Switched Arms
Description: HAQ-DI is a 20-question instrument that assesses the degree of difficulty of a participant in accomplishing tasks in eight functional areas: dressing and grooming, arising, eating, walking, hygiene, reach, grip and common daily activities. Overall HAQ-DI score was computed as sum of the domain scores divided by the number of domains answered. The total possible score ranges from 0 to 3 where 0 = least difficulty and 3 = extreme difficulty. Higher overall score indicates greater disability. A negative change from baseline indicates an improvement. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For efficacy assessments baseline is interpreted as Day 1.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo + MTX and GSK3196165 90mg + MTX | Placebo + MTX and GSK3196165 150mg + MTX | Placebo + MTX and Tofacitinib 5mg + MTX
Number analyzed (Participants) | 85 | 86 | 85
Scores on a scale
  Week 24 | -0.53 (0.065) | -0.46 (0.062) | -0.58 (0.062)
  Week 52 | -0.47 (0.069) | -0.45 (0.066) | -0.67 (0.065)

45. Secondary Outcome: Change From Baseline in Arthritis Pain VAS at Week 12
Description: For the Arthritis Pain VAS, participants assess the severity of their current arthritis pain using a continuous visual analogue scale (VAS) with anchors at "0" (no pain) and "100" (most severe pain). A negative change from baseline indicates an improvement. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX | Pooled Placebo
Number analyzed (Participants) | 513 | 510 | 258 | 256
Scores on a scale | -22 (1.056) | -19.56 (1.033) | -27.26 (1.473) | -14.58 (1.466)

46. Secondary Outcome: Change From Baseline in Arthritis Pain VAS at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1
Description: For the Arthritis Pain VAS, participants assess the severity of their current arthritis pain using a continuous visual analogue scale (VAS) with anchors at "0" (no pain) and "100" (most severe pain). A negative change from baseline indicates an improvement. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX
Number analyzed (Participants) | 513 | 510 | 258
Scores on a scale
  Week 24 | -25.43 (1.096) | -22.56 (1.069) | -31.02 (1.53)
  Week 52 | -28.36 (1.188) | -25.22 (1.175) | -33.34 (1.646)

47. Secondary Outcome: Change From Baseline in Arthritis Pain VAS at Week 24 and Week 52 for Placebo Switched Arms
Description: For the Arthritis Pain VAS, participants assess the severity of their current arthritis pain using a continuous visual analogue scale (VAS) with anchors at "0" (no pain) and "100" (most severe pain). A negative change from baseline indicates an improvement. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For efficacy assessments baseline is interpreted as Day 1.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo + MTX and GSK3196165 90mg + MTX | Placebo + MTX and GSK3196165 150mg + MTX | Placebo + MTX and Tofacitinib 5mg + MTX
Number analyzed (Participants) | 85 | 86 | 85
Scores on a scale
  Week 24 | -26.91 (2.666) | -28.02 (2.564) | -29.13 (2.566)
  Week 52 | -24.08 (2.902) | -29.22 (2.765) | -34.8 (2.742)

48. Secondary Outcome: Change From Baseline in Short Form (SF)-36 Physical Component Scores (PCS) at Week 12
Description: SF-36 is health-related survey that assesses quality of life covering 8 domains:physical functioning(PF),bodily pain(BP),role limitations due to physical/emotional problems,general health(GH),mental health,social functioning,vitality.Each of 8 domains is scored using average, 0-100; higher score represents better health.PCS was aggregated across the domains and scaled to T-score with mean of 50 and SD of 10; higher score represents better health.PCS is primarily derived from 4 domains(PF,role-physical,BP,GH) representing overall physical health.Positive change from baseline, reported using T-score change, indicates improvement in overall physical health.Quality Metric software was used for scoring.Baseline=latest pre-dose assessment with NMV, including those from unscheduled visits.CB=subtracting PD visit value from BV.For purpose of all analyses up to week12, placebo arms were pooled into single arm to primarily serve as reference for comparison of active treatment arms.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: T-Score
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX | Pooled Placebo
Number analyzed (Participants) | 513 | 510 | 258 | 256
T-Score | 5.38 (0.305) | 4.96 (0.297) | 6.93 (0.427) | 3.19 (0.423)

49. Secondary Outcome: Change From Baseline in SF-36 Mental Component Scores (MCS) at Week 12
Description: SF-36 is health-related survey that assesses quality of life covering 8 domains:physical functioning,bodily pain,role limitations due to physical/emotional problems,general health,mental health(MH),social functioning(SF),vitality.Each of 8 domains is scored using average, 0-100; higher score represents better health.MCS was aggregated across the domains and scaled to T-score with mean of 50 and SD of 10; higher score represents better health. MCS is primarily derived from 4 domains (SF,vitality,MH,role-emotional) representing overall mental health.Positive change from baseline, reported using T-score change, indicates improvement in overall mental health.Quality Metric software was used for scoring.Baseline=latest pre-dose assessment with NMV, including those from unscheduled visits.CB=subtracting PD visit value from BV.For purpose of all analyses up to week12, placebo arms were pooled into single arm to primarily serve as reference for comparison of active treatment arms.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: T-Score
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX | Pooled Placebo
Number analyzed (Participants) | 513 | 510 | 258 | 256
T-Score | 2.88 (0.41) | 2.54 (0.399) | 4.04 (0.574) | 2.46 (0.569)

50. Secondary Outcome: Change From Baseline in SF-36 Domain Scores at Week 12
Description: Short-Form 36 (SF-36) is a health-related survey that assesses quality of life covering 8 domains: physical functioning, bodily pain, role limitations due to physical and emotional problems, general health, mental health, social functioning, vitality. The MCS consists of 4 domains (SF, vitality, MH, role-emotional) and PCS consists of 4 domains (PF, role-physical, BP and GH).The individual question items are first summed for each item under the various sections. Then, those domain scores are weighted to a scale between 0 to 100, where higher score represents better health. A positive change from baseline indicates an improvement. Quality Metric software was used for scoring of SF-36.Baseline=latest pre-dose assessment with NMV, including those from unscheduled visits. CB=subtracting PD visit value from BV. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 28
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX | Pooled Placebo
Number analyzed (Participants) | 474 | 483 | 235 | 238
Scores on a scale
  Bodily Pain | 15.21 (21.448) | 14.65 (21.208) | 20.83 (22.432) | 10.39 (20.259)
  General Health | 8.23 (15.662) | 7.32 (15.462) | 11.11 (16.447) | 3.95 (14.251)
  Mental Health | 7.03 (18.222) | 6.4 (18.993) | 10.19 (18.659) | 4.35 (17.256)
  Physical Function | 13.2 (21.092) | 12.9 (21.564) | 17.81 (19.957) | 10.65 (22.363)
  Role Emotional | 7.47 (25.231) | 7.35 (25.162) | 9.25 (25.836) | 8.19 (24.699)
  Role Physical | 12.51 (21.751) | 12.56 (23.345) | 16.28 (22.117) | 8.8 (21.241)
  Social Function | 9.2 (23.558) | 8.72 (26.227) | 14.15 (25.092) | 8.98 (23.869)
  Vitality | 11.05 (20.216) | 9.82 (19.662) | 14.63 (20.185) | 8.14 (17.855)

51. Secondary Outcome: Change From Baseline in SF-36 PCS at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1
Description: SF-36 is health-related survey that assesses quality of life covering 8 domains:physical functioning(PF),bodily pain(BP),role limitations due to physical/emotional problems,general health(GH),mental health,social functioning,vitality.Each of 8 domains is scored using average, 0-100; higher score represents better health.PCS was aggregated across the domains and scaled to T-score with mean of 50 and SD of 10; higher score represents better health.PCS is primarily derived from 4 domains(PF,role-physical,BP,GH) representing overall physical health.Positive change from baseline, reported using T-score change, indicates improvement in overall physical health.Quality Metric software was used for scoring. Baseline was defined as latest pre-dose assessment with non-missing value, including from unscheduled visits. Change from Baseline was calculated by subtracting post dose visit value from Baseline value.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: T-Score
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX
Number analyzed (Participants) | 513 | 510 | 258
T-Score
  Week 24 | 6.26 (0.319) | 5.82 (0.313) | 8.07 (0.448)
  Week 52 | 6.5 (0.364) | 6.04 (0.358) | 8.23 (0.507)

52. Secondary Outcome: Change From Baseline in SF-36 MCS at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1
Description: SF-36 is health-related survey that assesses quality of life covering 8 domains:physical functioning,bodily pain,role limitations due to physical/emotional problems,general health,mental health(MH),social functioning(SF),vitality.Each of 8 domains is scored using average, 0-100; higher score represents better health.MCS was aggregated across the domains and scaled to T-score with mean of 50 and SD of 10; higher score represents better health. MCS is primarily derived from 4 domains (SF,vitality,MH,role-emotional) representing overall mental health.Positive change from baseline, reported using T-score change, indicates improvement in overall mental health.Quality Metric software was used for scoring. Baseline was defined as latest pre-dose assessment with non-missing value, including from unscheduled visits. Change from Baseline was calculated by subtracting post dose visit value from Baseline value.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: T-Score
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX
Number analyzed (Participants) | 513 | 510 | 258
T-Score
  Week 24 | 3.69 (0.401) | 3.87 (0.393) | 2.92 (0.563)
  Week 52 | 3.13 (0.443) | 2.75 (0.437) | 3.53 (0.616)

53. Secondary Outcome: Change From Baseline in SF-36 Domain Scores at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1
Description: The Short-Form 36 (SF-36) is a health-related survey that assesses quality of life covering 8 domains: physical functioning, bodily pain, role limitations due to physical and emotional problems, general health, mental health, social functioning, vitality. The MCS consists of 4 domains (social functioning, vitality, mental health, and role-emotional domains) and PCS consists of 4 domains (physical functioning, role-physical, bodily pain and general health). The individual question items are first summed for each item under the various sections. Then, those domain scores are weighted to a scale between 0 to 100, where higher score represents better health. A positive change from baseline indicates an improvement. Quality Metric software was used for scoring for SF-36. Baseline was defined as latest pre-dose assessment with non-missing value, including from unscheduled visits. Change from Baseline was calculated by subtracting post dose visit value from Baseline value.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 29
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX
Number analyzed (Participants) | 459 | 469 | 227
Scores on a scale
  Bodily Pain, Week 24 | 18.8 (21.717) | 18.06 (21.303) | 23.07 (22.7)
  Bodily Pain, Week 52: number analyzed (Participants) | 433 | 439 | 215
  Bodily Pain, Week 52 | 18.93 (23.084) | 18.39 (22.667) | 24.87 (23.427)
  General Health, Week 24 | 9.7 (15.747) | 9.01 (15.577) | 11.46 (16.416)
  General Health, Week 52: number analyzed (Participants) | 433 | 439 | 215
  General Health, Week 52 | 10.2 (16.795) | 8.81 (17.426) | 12.4 (19.371)
  Mental Health, Week 24 | 9.14 (17.511) | 8.88 (19.515) | 9.89 (18.461)
  Mental Health, Week 52: number analyzed (Participants) | 433 | 439 | 215
  Mental Health, Week 52 | 8.65 (18.468) | 7.43 (20.048) | 10.44 (21.685)
  Physical Function, Week 24 | 16.35 (22.51) | 16.2 (23.122) | 20.9 (21.808)
  Physical Function, Week 52: number analyzed (Participants) | 433 | 439 | 215
  Physical Function, Week 52 | 16.18 (24.737) | 17.22 (23.464) | 21.77 (25.534)
  Role Emotional, Week 24 | 10.75 (25.123) | 10.54 (25.451) | 7.86 (25.124)
  Role Emotional, Week 52: number analyzed (Participants) | 433 | 439 | 215
  Role Emotional, Week 52 | 10.08 (26.113) | 9.24 (26.689) | 9.3 (26.279)
  Role Physical, Week 24 | 15.35 (22.432) | 14.87 (23.361) | 18.81 (22.588)
  Role Physical, Week 52: number analyzed (Participants) | 433 | 439 | 215
  Role Physical, Week 52 | 16.5 (23.981) | 14.74 (24.325) | 19.16 (24.391)
  Social Function, Week 24 | 11.6 (23.543) | 12.95 (26.72) | 13.49 (24.164)
  Social Function, Week 52: number analyzed (Participants) | 433 | 439 | 215
  Social Function, Week 52 | 11.66 (25.523) | 10.51 (26.367) | 15.29 (24.872)
  Vitality, Week 24 | 13.37 (19.908) | 13.02 (20.115) | 15.5 (19.854)
  Vitality, Week 52: number analyzed (Participants) | 433 | 439 | 215
  Vitality, Week 52 | 13.37 (20.358) | 12.23 (20.712) | 15.73 (21.767)

54. Secondary Outcome: Change From Baseline in SF-36 PCS at Week 24 and Week 52 for Placebo Switched Arms
Description: SF-36 is health-related survey that assesses quality of life covering 8 domains:physical functioning(PF),bodily pain(BP),role limitations due to physical/emotional problems,general health(GH),mental health,social functioning,vitality. Each of 8 domains is scored using average, 0-100; higher score represents better health. PCS was aggregated across the domains and scaled to T-score with mean of 50 and SD of 10; higher score represents better health. PCS is primarily derived from 4 domains (PF,role-physical,BP,GH) representing overall physical health. Positive change from baseline, reported using T-score change, indicates improvement in overall physical health. Quality Metric software was used for scoring. Baseline was defined as latest pre-dose assessment with non-missing value, including from unscheduled visits. Change from Baseline was calculated by subtracting post dose visit value from Baseline value. For efficacy assessments baseline is interpreted as Day 1.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: T-Score
Arm/Group | Placebo + MTX and GSK3196165 90mg + MTX | Placebo + MTX and GSK3196165 150mg + MTX | Placebo + MTX and Tofacitinib 5mg + MTX
Number analyzed (Participants) | 85 | 86 | 85
T-Score
  Week 24 | 6.31 (0.773) | 7.07 (0.746) | 8.21 (0.747)
  Week 52 | 5.68 (0.89) | 6.27 (0.852) | 8.81 (0.848)

55. Secondary Outcome: Change From Baseline in SF-36 MCS at Week 24 and Week 52 for Placebo Switched Arms
Description: SF-36 is health-related survey that assesses quality of life covering 8 domains:physical functioning,bodily pain,role limitations due to physical/emotional problems,general health,mental health(MH),social functioning(SF),vitality. Each of 8 domains is scored using average, 0-100; higher score represents better health. MCS was aggregated across the domains and scaled to T-score with mean of 50 and SD of 10; higher score represents better health. MCS is primarily derived from 4 domains (SF,vitality,MH,role-emotional) representing overall mental health. Positive change from baseline, reported using T-score change, indicates improvement in overall mental health. Quality Metric software was used for scoring. Baseline was defined as latest pre-dose assessment with non-missing value, including from unscheduled visits. Change from Baseline was calculated by subtracting post dose visit value from Baseline value. For efficacy assessments baseline is interpreted as Day 1.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: T-Score
Arm/Group | Placebo + MTX and GSK3196165 90mg + MTX | Placebo + MTX and GSK3196165 150mg + MTX | Placebo + MTX and Tofacitinib 5mg + MTX
Number analyzed (Participants) | 85 | 86 | 85
T-Score
  Week 24 | 3.76 (0.973) | 4.43 (0.938) | 4.2 (0.942)
  Week 52 | 3.06 (1.081) | 3.77 (1.032) | 5.47 (1.027)

56. Secondary Outcome: Change From Baseline in SF-36 Domain Scores at Week 24 and Week 52 for Placebo Switched Arms
Description: Short-Form 36 (SF-36) is a health-related survey that assesses quality of life covering 8 domains: physical functioning(PF), bodily pain(BP), role limitations due to physical and emotional problems, general health(GH), mental health(MH), social functioning(SF), vitality. The MCS consists of 4 domains (SF, vitality, MH, role-emotional) and PCS consists of 4 domains (PF, role-physical, BP, GH). The individual question items are first summed for each item under the various sections. Then, those domain scores are weighted to a scale between 0 to 100, where higher score represents better health. A positive change from baseline indicates an improvement. Quality Metric software was used for scoring for SF-36. Baseline was defined as latest pre-dose assessment with non-missing value, including from unscheduled visits. Change from Baseline was calculated by subtracting post dose visit value from Baseline value. For efficacy assessments baseline is interpreted as Day 1.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 30
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo + MTX and GSK3196165 90mg + MTX | Placebo + MTX and GSK3196165 150mg + MTX | Placebo + MTX and Tofacitinib 5mg + MTX
Number analyzed (Participants) | 75 | 81 | 80
Scores on a scale
  Bodily Pain, Week 24 | 20.13 (23.373) | 23.28 (20.682) | 22.23 (20.389)
  Bodily Pain, Week 52: number analyzed (Participants) | 67 | 75 | 76
  Bodily Pain, Week 52 | 21.00 (24.696) | 24.96 (22.495) | 26.68 (22.838)
  General Health, Week 24 | 9.6 (18.212) | 12.02 (15.209) | 9.44 (13.61)
  General Health, Week 52: number analyzed (Participants) | 67 | 75 | 76
  General Health, Week 52 | 9.46 (16.95) | 9.00 (15.591) | 9.38 (15.469)
  Mental Health, Week 24 | 8.67 (18.405) | 9.81 (16.21) | 6.94 (16.41)
  Mental Health, Week 52: number analyzed (Participants) | 67 | 75 | 76
  Mental Health, Week 52 | 9.55 (22.271) | 9.87 (18.214) | 9.14 (17.576)
  Physical Function, Week 24 | 18.2 (20.725) | 21.42 (24.94) | 20.69 (22.385)
  Physical Function, Week 52: number analyzed (Participants) | 67 | 75 | 76
  Physical Function, Week 52 | 15.6 (25.13) | 18.87 (26.655) | 22.89 (20.22)
  Role Emotional, Week 24 | 12.89 (27.478) | 14.71 (24.73) | 10.83 (26.131)
  Role Emotional, Week 52: number analyzed (Participants) | 67 | 75 | 76
  Role Emotional, Week 52 | 10.07 (28.705) | 13.11 (29.612) | 13.92 (28.231)
  Role Physical, Week 24 | 17.83 (24.739) | 17.36 (24.065) | 17.58 (19.053)
  Role Physical, Week 52: number analyzed (Participants) | 67 | 75 | 76
  Role Physical, Week 52 | 18.38 (25.35) | 17.08 (26.443) | 21.05 (19.144)
  Social Function, Week 24 | 16.83 (21.503) | 16.36 (22.504) | 15.47 (23.804)
  Social Function, Week 52: number analyzed (Participants) | 67 | 75 | 76
  Social Function, Week 52 | 16.6 (25.505) | 14.00 (25.165) | 20.56 (25.389)
  Vitality, Week 24 | 15.92 (19.176) | 18.36 (19.196) | 15.31 (17.731)
  Vitality, Week 52: number analyzed (Participants) | 67 | 75 | 76
  Vitality, Week 52 | 16.14 (19.769) | 16.42 (17.671) | 16.12 (19.345)

57. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue at Week 12
Description: The Functional Assessment of Chronic Illness Therapy (FACIT)-fatigue is a validated patient-reported measure of 13 statements regarding the feeling of fatigue. The total score ranges from 0 to 52 with higher values representing a lower fatigue and a better quality of life. A positive change from baseline in FACIT-fatigue indicates an improvement. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX | Pooled Placebo
Number analyzed (Participants) | 513 | 510 | 258 | 256
Scores on a scale | 7.07 (0.41) | 6.3 (0.399) | 8.28 (0.577) | 4.72 (0.57)

58. Secondary Outcome: Change From Baseline in FACIT-Fatigue at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1
Description: The Functional Assessment of Chronic Illness Therapy (FACIT)-fatigue is a validated patient-reported measure of 13 statements regarding the feeling of fatigue. The total score ranges from 0 to 52 with higher values representing a lower fatigue and a better quality of life. A positive change from baseline in FACIT-fatigue indicates an improvement. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX
Number analyzed (Participants) | 513 | 510 | 258
Scores on a scale
  Week 24 | 8.52 (0.418) | 7.59 (0.406) | 8.56 (0.585)
  Week 52 | 7.71 (0.453) | 6.76 (0.446) | 8.55 (0.632)

59. Secondary Outcome: Change From Baseline in FACIT-Fatigue at Week 24 and Week 52 for Placebo Switched Arms
Description: The Functional Assessment of Chronic Illness Therapy (FACIT)-fatigue is a validated patient-reported measure of 13 statements regarding the feeling of fatigue. The total score ranges from 0 to 52 with higher values representing a lower fatigue and a better quality of life. A positive change from baseline in FACIT-fatigue indicates an improvement. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For efficacy assessments baseline is interpreted as Day 1.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo + MTX and GSK3196165 90mg + MTX | Placebo + MTX and GSK3196165 150mg + MTX | Placebo + MTX and Tofacitinib 5mg + MTX
Number analyzed (Participants) | 85 | 86 | 85
Scores on a scale
  Week 24 | 7.57 (1.002) | 7.91 (0.965) | 9.44 (0.969)
  Week 52 | 7.08 (1.102) | 7.2 (1.051) | 11.05 (1.043)

60. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESI)
Description: An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. SAEs are defined as any untoward medical occurrence that, at any dose: results in death, cause life threatening events which requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability or incapacity and birth defect or congenital anomaly. Protocol defined AESIs were included. Fifteen participants in Pooled placebo group who received active treatment of Tofacitinib from Week 4 instead of Week 12 as planned. They were pooled with the Tofacitinib arm in safety analysis.
Time Frame: Up to Week 59
Population: The analysis was performed on the Safety Set for Pooled Placebo (collected data till Week 12), GSK3196165 90 mg + MTX, GSK3196165 150 mg + MTX, Tofacitinib 5 mg + MTX (collected data till Week 59).
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX | Pooled Placebo
Number analyzed (Participants) | 513 | 510 | 273 | 241
Participants
  Participants with AE | 367 | 383 | 207 | 95
  Participants with SAE | 33 | 39 | 23 | 8
  Participants with AESI | 65 | 58 | 22 | 4

61. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESI) for Placebo Switched Arms
Description: An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. SAEs are defined as any untoward medical occurrence that, at any dose: results in death, cause life threatening events which requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability or incapacity and birth defect or congenital anomaly. Protocol defined AESIs were included.
Time Frame: Up to Week 59
Population: The analysis was performed on Safety Set-Placebo switch for Placebo + MTX and GSK3196165 90 mg + MTX, Placebo + MTX and GSK3196165 150 mg + MTX, Placebo + MTX and Tofacitinib 5 mg + MTX (collected data from Week 12 to 59).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + MTX and GSK3196165 90mg + MTX | Placebo + MTX and GSK3196165 150mg + MTX | Placebo + MTX and Tofacitinib 5mg + MTX
Number analyzed (Participants) | 80 | 82 | 68
Participants
  Participants with AE | 49 | 52 | 44
  Participants with SAE | 8 | 9 | 5
  Participants with AESI | 9 | 9 | 3

62. Secondary Outcome: Change From Baseline in White Blood Cell (WBC) Count at Week 12
Description: Blood samples were collected for the assessment of hematology parameter white blood cell count. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 1) and Week 12
Population: The analysis was performed on the Safety Set. Fifteen participants in Pooled placebo group who received active treatment of Tofacitinib from Week 4 instead of Week 12 as planned. They were pooled with the Tofacitinib arm in safety analysis. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Giga cells per liter (10^9/L)
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX | Pooled Placebo
Number analyzed (Participants) | 456 | 455 | 230 | 213
Giga cells per liter (10^9/L) | -0.55 (2.267) | -0.63 (2.065) | -1.03 (2.16) | -0.3 (2.005)

63. Secondary Outcome: Change From Baseline in WBC Count at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1
Description: Blood samples were collected for the assessment of hematology parameter white blood cell count. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 62
Measure: Mean (Standard Deviation); unit: Giga cells per liter (10^9/L)
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX
Number analyzed (Participants) | 443 | 465 | 246
Giga cells per liter (10^9/L)
  Week 24 | -0.59 (2.279) | -0.5 (2.123) | -0.94 (2.31)
  Week 52: number analyzed (Participants) | 381 | 396 | 219
  Week 52 | -0.54 (2.386) | -0.52 (2.051) | -1.21 (2.407)

64. Secondary Outcome: Change From Baseline in WBC Count at Week 24 and Week 52 for Placebo Switched Arms
Description: Blood samples were collected for the assessment of hematology parameter white blood cell count. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For safety assessments baseline is interpreted as Week 12.
Time Frame: Baseline (Week 12), Week 24 and Week 52
Population: The analysis was performed on the Safety Set-Placebo switch. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Giga cells per liter (10^9/L)
Arm/Group | Placebo + MTX and GSK3196165 90mg + MTX | Placebo + MTX and GSK3196165 150mg + MTX | Placebo + MTX and Tofacitinib 5mg + MTX
Number analyzed (Participants) | 78 | 78 | 63
Giga cells per liter (10^9/L)
  Week 24 | -0.06 (1.94) | -0.31 (1.642) | -0.61 (2.052)
  Week 52: number analyzed (Participants) | 61 | 68 | 55
  Week 52 | -0.21 (2.129) | -0.03 (2.459) | -0.96 (2.013)

65. Secondary Outcome: Change From Baseline in Hematology Parameter of Platelet Count, Neutrophils, Lymphocytes at Week 12
Description: Blood samples were collected for the assessment of hematology parameters including platelet count, neutrophils, lymphocytes. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 62
Measure: Mean (Standard Deviation); unit: Giga cells per liter (10^9/L)
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX | Pooled Placebo
Number analyzed (Participants) | 453 | 454 | 229 | 211
Giga cells per liter (10^9/L)
  Lymphocytes: number analyzed (Participants) | 453 | 451 | 227 | 211
  Lymphocytes | 0.006 (0.5341) | 0.016 (0.5552) | 0.084 (0.5789) | -0.009 (0.5367)
  Neutrophils: number analyzed (Participants) | 453 | 451 | 227 | 211
  Neutrophils | -0.565 (2.2309) | -0.66 (2.0562) | -1.076 (2.162) | -0.268 (2.025)
  Platelets: number analyzed (Participants) | 452 | 454 | 229 | 211
  Platelets | -18.6 (58.93) | -16.3 (59.51) | -26.7 (63.56) | -1 (58.79)

66. Secondary Outcome: Change From Baseline in Hematology Parameter of Platelet Count, Neutrophils, Lymphocytes at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1
Description: Blood samples were collected for the assessment of hematology parameters including platelet count, neutrophils, lymphocytes. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 62
Measure: Mean (Standard Deviation); unit: Giga cells per liter (10^9/L)
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX
Number analyzed (Participants) | 442 | 464 | 246
Giga cells per liter (10^9/L)
  Lymphocytes, Week 24 | 0.031 (0.583) | -0.003 (0.5395) | 0.017 (0.62)
  Lymphocytes, Week 52: number analyzed (Participants) | 378 | 394 | 219
  Lymphocytes, Week 52 | 0.015 (0.5485) | -0.034 (0.5771) | -0.102 (0.5877)
  Neutrophils, Week 24 | -0.629 (2.2736) | -0.515 (1.9997) | -0.899 (2.2436)
  Neutrophils, Week 52: number analyzed (Participants) | 378 | 393 | 219
  Neutrophils, Week 52 | -0.583 (2.3708) | -0.493 (1.9958) | -1.049 (2.3054)
  Platelets, Week 24: number analyzed (Participants) | 442 | 464 | 245
  Platelets, Week 24 | -13.7 (65.69) | -15.4 (67.72) | -27.1 (70.17)
  Platelets, Week 52: number analyzed (Participants) | 376 | 391 | 217
  Platelets, Week 52 | -18.7 (66.07) | -18.5 (64.59) | -30.2 (56.67)

67. Secondary Outcome: Change From Baseline in Hematology Parameter of Platelet Count, Neutrophils, Lymphocytes at Week 24 and Week 52 for Placebo Switched Arms
Description: Blood samples were collected for the assessment of hematology parameters including platelet count, neutrophils, lymphocytes. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For safety assessments baseline is interpreted as Week 12.
Time Frame: Baseline (Week 12), Week 24 and Week 52
Population: as for outcome 64
Measure: Mean (Standard Deviation); unit: Giga cells per liter (10^9/L)
Arm/Group | Placebo + MTX and GSK3196165 90mg + MTX | Placebo + MTX and GSK3196165 150mg + MTX | Placebo + MTX and Tofacitinib 5mg + MTX
Number analyzed (Participants) | 78 | 78 | 63
Giga cells per liter (10^9/L)
  Lymphocytes, Week 24 | -0.055 (0.5751) | 0.038 (0.5294) | 0.085 (0.5052)
  Lymphocytes, Week 52: number analyzed (Participants) | 60 | 67 | 54
  Lymphocytes, Week 52 | -0.091 (0.6046) | 0.09 (0.5744) | -0.079 (0.4538)
  Neutrophils, Week 24 | -0.053 (1.8784) | -0.405 (1.5633) | -0.685 (1.9031)
  Neutrophils, Week 52: number analyzed (Participants) | 60 | 67 | 54
  Neutrophils, Week 52 | -0.118 (2.0773) | -0.289 (2.3914) | -0.847 (1.8472)
  Platelets, Week 24: number analyzed (Participants) | 77 | 76 | 63
  Platelets, Week 24 | -11.3 (59.64) | -17.4 (63.81) | -9.3 (43.83)
  Platelets, Week 52: number analyzed (Participants) | 60 | 67 | 55
  Platelets, Week 52 | -19 (65.35) | -11.7 (86.52) | -19.6 (51.16)

68. Secondary Outcome: Change From Baseline in Hematology Parameter of Hemoglobin at Week 12
Description: Blood samples were collected for the assessment of change from baseline in hematology parameters hemoglobin level. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 1) and Week 12
Population: The analysis was performed on the Safety Set participants. Fifteen participants in Pooled placebo group who received active treatment of Tofacitinib from Week 4 instead of Week 12 as planned. They were pooled with the Tofacitinib arm in safety analysis. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX | Pooled Placebo
Number analyzed (Participants) | 457 | 459 | 231 | 214
Grams per liter (g/L) | -0.0 (8.14) | 0.5 (8.5) | 0.0 (8.56) | -1.7 (7.83)

69. Secondary Outcome: Change From Baseline in Hematology Parameter of Hemoglobin at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1
Description: Blood samples were collected for the assessment of change from baseline in hematology parameters hemoglobin level. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 68
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX
Number analyzed (Participants) | 444 | 466 | 246
Grams per liter (g/L)
  Week 24 | 0.5 (8.96) | 1.3 (9.22) | 1.1 (9.23)
  Week 52: number analyzed (Participants) | 381 | 397 | 219
  Week 52 | 0.4 (9.5) | 0.7 (9.24) | -0.2 (9.14)

70. Secondary Outcome: Change From Baseline in Hematology Parameter of Hemoglobin at Week 24 and Week 52 for Placebo Switched Arms
Description: Blood samples were collected for the assessment of change from baseline in hematology parameters hemoglobin level. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For safety assessments baseline is interpreted as Week 12.
Time Frame: Baseline (Week 12), Week 24 and Week 52
Population: as for outcome 64
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | Placebo + MTX and GSK3196165 90mg + MTX | Placebo + MTX and GSK3196165 150mg + MTX | Placebo + MTX and Tofacitinib 5mg + MTX
Number analyzed (Participants) | 78 | 78 | 63
Grams per liter (g/L)
  Week 24 | 0.7 (8.72) | 2 (9.02) | 1.8 (6.71)
  Week 52: number analyzed (Participants) | 61 | 68 | 55
  Week 52 | 1.4 (9.85) | 1.1 (10.57) | 0.8 (8.81)

71. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter of Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Alkaline Phosphatase (AP), Gamma-Glutamyl Transpeptidase (GGT) at Week 12
Description: Blood samples were collected for the assessment of clinical chemistry parameters including aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (AP) and gamma-glutamyl transferase (GGT) levels. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 68
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX | Pooled Placebo
Number analyzed (Participants) | 468 | 475 | 242 | 220
International units per liter (IU/L)
  Alkaline Phosphatase | -1.5 (17.97) | -1.2 (15.64) | -3.7 (16.07) | -0.7 (15.29)
  ALT: number analyzed (Participants) | 467 | 475 | 242 | 220
  ALT | 0.5 (15.69) | 2 (19.66) | 2.2 (15.07) | -1.1 (11.76)
  AST: number analyzed (Participants) | 467 | 475 | 241 | 220
  AST | 1.2 (9.71) | 2.4 (13.09) | 3.1 (14.09) | -0.4 (7.38)
  Gamma Glutamyl Transferase | -2.1 (17.67) | -2.3 (16.05) | 1.2 (23.21) | -0.5 (16.31)

72. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter of AST, ALT, AP, GGT at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1
Description: Blood samples were collected for the assessment of clinical chemistry parameters including AST, ALT, AP and GGT levels. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 68
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX
Number analyzed (Participants) | 448 | 467 | 246
International units per liter (IU/L)
  Alkaline Phosphatase, Week 24 | 0.5 (17.77) | 1.8 (19.16) | -3.0 (17.41)
  Alkaline Phosphatase, Week 52: number analyzed (Participants) | 395 | 407 | 222
  Alkaline Phosphatase, Week 52 | 2.8 (19.52) | 1.5 (17.35) | -1.0 (18.12)
  ALT, Week 24 | 1.5 (22.98) | 2.5 (17.22) | 4.5 (40.51)
  ALT, Week 52: number analyzed (Participants) | 395 | 407 | 222
  ALT, Week 52 | 0.4 (12.31) | -0.2 (13.95) | 1.9 (15.72)
  AST, Week 24 | 1.3 (11.36) | 2.4 (11.25) | 8.6 (94.12)
  AST, Week 52: number analyzed (Participants) | 394 | 407 | 222
  AST, Week 52 | 1.0 (8.97) | 1.0 (8.22) | 3.1 (14.21)
  Gamma Glutamyl Transferase, Week 24: number analyzed (Participants) | 448 | 466 | 246
  Gamma Glutamyl Transferase, Week 24 | -1.7 (18.05) | -1.2 (17.71) | 0.2 (19.7)
  Gamma Glutamyl Transferase, Week 52: number analyzed (Participants) | 395 | 407 | 222
  Gamma Glutamyl Transferase, Week 52 | -0.3 (22.26) | -0.4 (22.03) | 1.6 (20.52)

73. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter of AST, ALT, AP, GGT at Week 24 and Week 52 for Placebo Switched Arms
Description: Blood samples were collected for the assessment of clinical chemistry parameters including AST, ALT, AP and GGT levels. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For safety assessments baseline is interpreted as Week 12.
Time Frame: Baseline (Week 12), Week 24 and Week 52
Population: as for outcome 64
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | Placebo + MTX and GSK3196165 90mg + MTX | Placebo + MTX and GSK3196165 150mg + MTX | Placebo + MTX and Tofacitinib 5mg + MTX
Number analyzed (Participants) | 78 | 78 | 63
International units per liter (IU/L)
  Alkaline Phosphatase, Week 24 | 0.9 (13.07) | -0.3 (18.04) | 0.7 (14.91)
  Alkaline Phosphatase, Week 52: number analyzed (Participants) | 65 | 72 | 58
  Alkaline Phosphatase, Week 52 | 5.5 (24.05) | -1.9 (16.07) | -1 (14.6)
  ALT, Week 24 | 0.3 (10.76) | 3.6 (18.43) | 3.3 (13.9)
  ALT, Week 52: number analyzed (Participants) | 65 | 72 | 58
  ALT, Week 52 | 2.6 (15.59) | 2.6 (11.55) | 2.7 (15.03)
  AST, Week 24 | 1.5 (11.4) | 2.9 (13.53) | 3.2 (10.53)
  AST, Week 52: number analyzed (Participants) | 65 | 72 | 58
  AST, Week 52 | 1.8 (6.89) | 2 (9.08) | 3.6 (9.88)
  Gamma Glutamyl Transferase, Week 24 | 0.8 (13.65) | 0.9 (16.68) | -0.5 (32.46)
  Gamma Glutamyl Transferase, Week 52: number analyzed (Participants) | 65 | 72 | 58
  Gamma Glutamyl Transferase, Week 52 | 8.1 (55.51) | 1 (14.4) | -2.2 (35.14)

74. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter of Total Bilirubin at Week 12
Description: Blood samples were collected for the assessment of clinical chemistry parameter total bilirubin level. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 68
Measure: Mean (Standard Deviation); unit: Micromoles per liter (umol/L)
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX | Pooled Placebo
Number analyzed (Participants) | 468 | 475 | 242 | 220
Micromoles per liter (umol/L) | 0.3 (2.63) | 0.4 (2.52) | 0.5 (2.96) | -0.2 (3.13)

75. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter of Total Bilirubin at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1
Description: Blood samples were collected for the assessment of clinical chemistry parameter total bilirubin level. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 68
Measure: Mean (Standard Deviation); unit: Micromoles per liter (umol/L)
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX
Number analyzed (Participants) | 448 | 467 | 246
Micromoles per liter (umol/L)
  Week 24 | 0.5 (2.93) | 0.6 (2.79) | 0.6 (2.95)
  Week 52: number analyzed (Participants) | 395 | 408 | 222
  Week 52 | 0.5 (2.73) | 0.4 (2.81) | 0.5 (3.2)

76. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter of Total Bilirubin at Week 24 and Week 52 for Placebo Switched Arms
Description: Blood samples were collected for the assessment of clinical chemistry parameter total bilirubin level. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For safety assessments baseline is interpreted as Week 12.
Time Frame: Baseline (Week 12), Week 24 and Week 52
Population: as for outcome 64
Measure: Mean (Standard Deviation); unit: Micromoles per liter (umol/L)
Arm/Group | Placebo + MTX and GSK3196165 90mg + MTX | Placebo + MTX and GSK3196165 150mg + MTX | Placebo + MTX and Tofacitinib 5mg + MTX
Number analyzed (Participants) | 78 | 78 | 63
Micromoles per liter (umol/L)
  Week 24 | 0.2 (2.65) | 0.6 (2.8) | 0.1 (2.62)
  Week 52: number analyzed (Participants) | 65 | 72 | 58
  Week 52 | 0.3 (3.16) | 0.6 (2.75) | 0.6 (2.64)

77. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter of Albumin at Week 12
Description: Blood samples were collected for the assessment of clinical chemistry parameter albumin level. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 68
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX | Pooled Placebo
Number analyzed (Participants) | 468 | 475 | 242 | 220
Grams per liter (g/L) | -0.2 (2.7) | 0.2 (2.53) | 0.8 (3.05) | -0.7 (2.7)

78. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter of Albumin at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1
Description: Blood samples were collected for the assessment of clinical chemistry parameter albumin level. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 68
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX
Number analyzed (Participants) | 448 | 466 | 246
Grams per liter (g/L)
  Week 24 | 0.2 (2.85) | 0.3 (2.69) | 1.3 (3.17)
  Week 52: number analyzed (Participants) | 395 | 408 | 222
  Week 52 | -0.2 (3.08) | 0.3 (3.03) | 0.6 (2.83)

79. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter of Albumin at Week 24 and Week 52 for Placebo Switched Arms
Description: Blood samples were collected for the assessment of clinical chemistry parameter albumin level. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For safety assessments baseline is interpreted as Week 12.
Time Frame: Baseline (Week 12), Week 24 and Week 52
Population: as for outcome 64
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | Placebo + MTX and GSK3196165 90mg + MTX | Placebo + MTX and GSK3196165 150mg + MTX | Placebo + MTX and Tofacitinib 5mg + MTX
Number analyzed (Participants) | 78 | 78 | 63
Grams per liter (g/L)
  Week 24 | 0.3 (2.57) | 1.1 (2.54) | 1.8 (2.47)
  Week 52: number analyzed (Participants) | 65 | 72 | 58
  Week 52 | 0.3 (2.94) | 0.8 (2.77) | 1.2 (2.24)

80. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of Total Cholesterol at Week 12
Description: Blood samples were collected for the assessment of lipid profile of total cholesterol levels. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 1) and Week 12
Population: Blood samples were collected at indicated time points per schedule of activities in protocol. Objectives and Endpoints section incorrectly states that Change from baseline in key laboratory parameters at Week 12 was a secondary objective, however for lipid profile, there is no corresponding time point in schedule of activities. Consequently, the objective cannot be assessed at the specified time points since the sample was collected at Week 4. Week 4 is not pre-specified time point to report.
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX | Pooled Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

81. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of Total Cholesterol at Week 24 for Treatment Arms Who Started Study Intervention From Day 1
Description: Blood samples were collected for the assessment of lipid profile of total cholesterol levels. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline (Day 1) and Week 24
Population: Blood samples were collected at indicated time points per schedule of activities in protocol. Objectives and Endpoints section incorrectly states that Change from baseline in key laboratory parameters at Week 24 was a secondary objective, however for lipid profile, there is no corresponding time point in schedule of activities. Consequently, the objective cannot be assessed at the specified time points since the sample was collected at Week 16. Week 16 is not pre-specified time point to report.
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX
Number analyzed (Participants) | 0 | 0 | 0

82. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of Total Cholesterol at Week 24 for Placebo Switched Arms
Description: Blood samples were collected for the assessment of lipid profile of total cholesterol levels. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For safety assessments baseline is interpreted as Week 12.
Time Frame: Baseline (Day 1) and Week 24
Population: as for outcome 81
Arm/Group | Placebo + MTX and GSK3196165 90mg + MTX | Placebo + MTX and GSK3196165 150mg + MTX | Placebo + MTX and Tofacitinib 5mg + MTX
Number analyzed (Participants) | 0 | 0 | 0

83. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of Total Cholesterol at Week 52 for Treatment Arms Who Started Study Intervention From Day 1
Description: as for outcome 81
Time Frame: Baseline (Day 1) and Week 52
Population: as for outcome 68
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX
Number analyzed (Participants) | 394 | 405 | 223
Millimoles per liter (mmol/L) | 0.084 (0.846) | 0.074 (0.9528) | 0.535 (0.9012)

84. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of Total Cholesterol at Week 52 for Placebo Switched Arms
Description: as for outcome 82
Time Frame: Baseline (Day 1) and Week 52
Population: as for outcome 64
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Placebo + MTX and GSK3196165 90mg + MTX | Placebo + MTX and GSK3196165 150mg + MTX | Placebo + MTX and Tofacitinib 5mg + MTX
Number analyzed (Participants) | 62 | 69 | 56
Millimoles per liter (mmol/L) | 0.334 (0.7608) | 0.045 (0.7931) | 0.486 (0.8974)

85. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of Low-density Lipoprotein (LDL) Cholesterol, High-density Lipoprotein-cholesterol at Week 12
Description: Blood samples were collected for the assessment of fasting lipid profile including LDL cholesterol, HDL cholesterol levels. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 80
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX | Pooled Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

86. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of LDL Cholesterol, High-density Lipoprotein-cholesterol at Week 24 for Treatment Arms Who Started Study Intervention From Day 1
Description: Blood samples were collected for the assessment of fasting lipid profile including LDL cholesterol, HDL cholesterol levels. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline (Day 1) and Week 24
Population: as for outcome 81
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX
Number analyzed (Participants) | 0 | 0 | 0

87. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of LDL Cholesterol, High-density Lipoprotein-cholesterol at Week 24 for Placebo Switched Arms
Description: Blood samples were collected for the assessment of fasting lipid profile including LDL cholesterol, HDL cholesterol levels. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For safety assessments baseline is interpreted as Week 12.
Time Frame: Baseline (Day 1) and Week 24
Population: as for outcome 81
Arm/Group | Placebo + MTX and GSK3196165 90mg + MTX | Placebo + MTX and GSK3196165 150mg + MTX | Placebo + MTX and Tofacitinib 5mg + MTX
Number analyzed (Participants) | 0 | 0 | 0

88. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of LDL Cholesterol, High-density Lipoprotein-cholesterol at Week 52 for Treatment Arms Who Started Study Intervention From Day 1
Description: as for outcome 86
Time Frame: Baseline (Day 1) and Week 52
Population: as for outcome 68
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX
Number analyzed (Participants) | 394 | 405 | 223
Millimoles per liter (mmol/L)
  HDL Cholesterol, Direct | -0.046 (0.3024) | 0.011 (0.2887) | 0.117 (0.2986)
  LDL Cholesterol: number analyzed (Participants) | 391 | 401 | 220
  LDL Cholesterol | 0.089 (0.7062) | 0.053 (0.736) | 0.369 (0.758)

89. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of LDL Cholesterol, High-density Lipoprotein-cholesterol at Week 52 for Placebo Switched Arms
Description: as for outcome 87
Time Frame: Baseline (Day 1) and Week 52
Population: as for outcome 64
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Placebo + MTX and GSK3196165 90mg + MTX | Placebo + MTX and GSK3196165 150mg + MTX | Placebo + MTX and Tofacitinib 5mg + MTX
Number analyzed (Participants) | 62 | 69 | 56
Millimoles per liter (mmol/L)
  HDL Cholesterol, Direct | 0.083 (0.302) | 0.033 (0.209) | 0.092 (0.2701)
  LDL Cholesterol: number analyzed (Participants) | 62 | 68 | 55
  LDL Cholesterol | 0.221 (0.6669) | -0.003 (0.697) | 0.304 (0.8315)

90. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of Triglycerides at Week 12
Description: Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 80
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX | Pooled Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

91. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of Triglycerides at Week 24 for Treatment Arms Who Started Study Intervention From Day 1
Description: Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline (Day 1) and Week 24
Population: as for outcome 81
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX
Number analyzed (Participants) | 0 | 0 | 0

92. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of Triglycerides at Week 24 for Placebo Switched Arms
Description: Blood samples were collected for the assessment of fasting lipid profile including triglycerides. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For safety assessments baseline is interpreted as Week 12.
Time Frame: Baseline (Day 1) and Week 24
Population: as for outcome 81
Arm/Group | Placebo + MTX and GSK3196165 90mg + MTX | Placebo + MTX and GSK3196165 150mg + MTX | Placebo + MTX and Tofacitinib 5mg + MTX
Number analyzed (Participants) | 0 | 0 | 0

93. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of Triglycerides at Week 52 for Treatment Arms Who Started Study Intervention From Day 1
Description: as for outcome 91
Time Frame: Baseline (Day 1) and Week 52
Population: as for outcome 68
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX
Number analyzed (Participants) | 394 | 405 | 223
Millimoles per liter (mmol/L) | 0.081 (0.5531) | 0.051 (0.7413) | 0.119 (0.7325)

94. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of Triglycerides at Week 52 for Placebo Switched Arms
Description: as for outcome 92
Time Frame: Baseline (Day 1) and Week 52
Population: as for outcome 64
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Placebo + MTX and GSK3196165 90mg + MTX | Placebo + MTX and GSK3196165 150mg + MTX | Placebo + MTX and Tofacitinib 5mg + MTX
Number analyzed (Participants) | 62 | 69 | 56
Millimoles per liter (mmol/L) | 0.066 (0.5071) | 0.03 (0.6306) | 0.241 (0.5357)

95. Secondary Outcome: Number of Participants With National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) >=Grade 3 Hematological/Clinical Chemistry Abnormalities
Description: Number of participants with NCI-CTCAE >=Grade 3 hematological/clinical chemistry abnormalities were summarized. Hematological and Clinical chemistry parameters were summarized according to the NCI-CTCAE, version 5.0: Grade 1: mild; Grade 2: moderate; Grade 3: severe; Grade 4: life-threatening or disabling. Higher grade indicates more severity. Data is presented for only those parameters for which participants had worst case >=Grade 3 shifts from Baseline. Fifteen participants in Pooled placebo group who received active treatment of Tofacitinib from Week 4 instead of Week 12 as planned. They were pooled with the Tofacitinib arm in safety analysis.
Time Frame: Up to Week 59
Population: as for outcome 60
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX | Pooled Placebo
Number analyzed (Participants) | 513 | 510 | 273 | 238
Participants
  Aspartate aminotransferase increased, Total, Grade 3: number analyzed (Participants) | 509 | 508 | 273 | 237
  Aspartate aminotransferase increased, Total, Grade 3 | 0 | 5 | 1 | 0
  Aspartate aminotransferase increased, Total, Grade 4: number analyzed (Participants) | 509 | 508 | 273 | 237
  Aspartate aminotransferase increased, Total, Grade 4 | 0 | 0 | 1 | 0
  Hypertriglyceridemia, Total, Grade 3: number analyzed (Participants) | 503 | 504 | 266 | 228
  Hypertriglyceridemia, Total, Grade 3 | 2 | 1 | 2 | 1
  Hypertriglyceridemia, Total, Grade 4: number analyzed (Participants) | 503 | 504 | 266 | 228
  Hypertriglyceridemia, Total, Grade 4 | 1 | 1 | 0 | 0
  Alanine aminotransferase increased, Total, Grade 3: number analyzed (Participants) | 509 | 508 | 273 | 237
  Alanine aminotransferase increased, Total, Grade 3 | 5 | 6 | 1 | 0
  Alanine aminotransferase increased, Total, Grade 4: number analyzed (Participants) | 509 | 508 | 273 | 237
  Alanine aminotransferase increased, Total, Grade 4 | 0 | 1 | 0 | 0
  Blood bilirubin increased, Total, Grade 3: number analyzed (Participants) | 509 | 508 | 273 | 237
  Blood bilirubin increased, Total, Grade 3 | 0 | 1 | 0 | 0
  Cholesterol - high, Total, Grade 3: number analyzed (Participants) | 503 | 504 | 266 | 228
  Cholesterol - high, Total, Grade 3 | 0 | 1 | 0 | 0
  Creatinine increased, Total, Grade 3: number analyzed (Participants) | 509 | 508 | 273 | 238
  Creatinine increased, Total, Grade 3 | 0 | 1 | 0 | 0
  Chronic Kidney Disease, Total Grade 3: number analyzed (Participants) | 509 | 508 | 273 | 238
  Chronic Kidney Disease, Total Grade 3 | 2 | 2 | 1 | 0
  Chronic Kidney Disease, Total Grade 4: number analyzed (Participants) | 509 | 508 | 273 | 238
  Chronic Kidney Disease, Total Grade 4 | 0 | 1 | 0 | 0
  Anemia, Total, Grade 3: number analyzed (Participants) | 509 | 508 | 273 | 237
  Anemia, Total, Grade 3 | 2 | 4 | 1 | 0
  White blood cell decreased, Total , Grade 3: number analyzed (Participants) | 509 | 508 | 273 | 237
  White blood cell decreased, Total , Grade 3 | 1 | 1 | 0 | 0
  Lymphocyte count decreased, Total, Grade 3: number analyzed (Participants) | 509 | 508 | 273 | 237
  Lymphocyte count decreased, Total, Grade 3 | 6 | 9 | 5 | 1
  Lymphocyte count decreased, Total, Grade 4: number analyzed (Participants) | 509 | 508 | 273 | 237
  Lymphocyte count decreased, Total, Grade 4 | 0 | 1 | 0 | 0
  Neutrophil count decreased, Total, Grade 3: number analyzed (Participants) | 509 | 508 | 273 | 237
  Neutrophil count decreased, Total, Grade 3 | 4 | 0 | 0 | 2
  Neutrophil count decreased, Total, Grade 4: number analyzed (Participants) | 509 | 508 | 273 | 237
  Neutrophil count decreased, Total, Grade 4 | 2 | 3 | 1 | 1
  Platelet count decreased, Total Grade 3: number analyzed (Participants) | 509 | 508 | 273 | 236
  Platelet count decreased, Total Grade 3 | 1 | 0 | 0 | 0
  Platelet count decreased, Total, Grade 4: number analyzed (Participants) | 509 | 508 | 273 | 236
  Platelet count decreased, Total, Grade 4 | 0 | 0 | 1 | 0

96. Secondary Outcome: Number of Participants With National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) >=Grade 3 Hematological/Clinical Chemistry Abnormalities for Placebo Switched Arms
Description: Number of participants with NCI-CTCAE >=Grade 3 hematological/clinical chemistry abnormalities were summarized. Hematological and Clinical chemistry parameters were summarized according to the NCI-CTCAE, version 5.0: Grade 1: mild; Grade 2: moderate; Grade 3: severe; Grade 4: life-threatening or disabling. Higher grade indicates more severity. Data is presented for only those parameters for which participants had worst case >=Grade 3 shifts from Baseline.
Time Frame: Up to Week 59
Population: as for outcome 61
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + MTX and GSK3196165 90mg + MTX | Placebo + MTX and GSK3196165 150mg + MTX | Placebo + MTX and Tofacitinib 5mg + MTX
Number analyzed (Participants) | 80 | 82 | 68
Participants
  Hypertriglyceridemia, Total, Grade 3 | 1 | 2 | 0
  Neutrophil count decreased, Grade 3, Grade 4 | 0 | 0 | 1
  Neutrophil count decreased, Grade 4, Grade 3 | 1 | 0 | 0
  Creatinine increased, Total, Grade 3 | 1 | 0 | 0
  Chronic Kidney Disease, Total Grade 3 | 2 | 0 | 0
  Anemia, Total, Grade 3 | 1 | 2 | 0
  White blood cell decreased, Total , Grade 3 | 1 | 0 | 0
  Lymphocyte count decreased, Total, Grade 3 | 0 | 0 | 1
  Lymphocyte count decreased, Total, Grade 4 | 0 | 1 | 0
  Neutrophil count decreased, Total, Grade 3 | 2 | 0 | 0
  Neutrophil count decreased, Total, Grade 4 | 0 | 0 | 2
  Platelet count decreased, Total Grade 3 | 0 | 0 | 1

97. Secondary Outcome: Concentrations of Granulocyte-macrophage Colony Stimulating Factor (GM-CSF) Autoantibody
Description: Concentrations of GM-CSF autoantibodies were determined.
Time Frame: At baseline
Population: The analysis was performed on the Safety Set. Fifteen participants in Pooled placebo group who received active treatment of Tofacitinib from Week 4 instead of Week 12 as planned. They were pooled with the Tofacitinib arm in safety analysis. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Microgram per liter (ug/L)
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX | Placebo + MTX and GSK3196165 90mg + MTX | Placebo + MTX and GSK3196165 150mg + MTX | Placebo + MTX and Tofacitinib 5mg + MTX
Number analyzed (Participants) | 491 | 486 | 264 | 82 | 85 | 70
Microgram per liter (ug/L) | 832.827 (12355.2805) | 218.456 (632.5733) | 203.31 (444.708) | 231.376 (446.1713) | 357.087 (629.3471) | 240.109 (624.4536)

98. Secondary Outcome: Number of Participants With Anti-GSK3196165 Antibodies
Description: Serum samples were collected for the determination of anti- GSK3196165 antibodies (ADA) using a validated electrochemiluminescence (ECL) immunoassay. The assay involved screening, confirmation and titration steps. If serum samples tested positive in the screening assay, they were considered 'potentially positive' and were further analyzed for the specificity using the confirmation assay. Samples that confirmed positive in the confirmation assay were reported as 'positive'. Confirmed positive ADA samples were further characterized in the titration assay to quasi-quantitate the amount of ADA in the sample. Additionally, confirmed positive ADA samples were also tested in a validated neutralizing antibody assay to determine the potential neutralizing activity of the ADA.
Time Frame: Up to Week 59
Population: as for outcome 97
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX | Placebo + MTX and GSK3196165 90mg + MTX | Placebo + MTX and GSK3196165 150mg + MTX | Placebo + MTX and Tofacitinib 5mg + MTX
Number analyzed (Participants) | 513 | 510 | 273 | 85 | 86 | 70
Participants | 7 | 7 | 0 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: All AEs and SAEs were collected from the start of study intervention. The Pooled Placebo collected during the timeframe Week 0 to Week 12. Placebo + MTX and GSK3196165 90 mg + MTX, Placebo + MTX and GSK3196165 150 mg + MTX, Placebo + MTX and Tofacitinib 5mg + MTX collected during the timeframe Week 12 to Week 59. GSK3196165 90 mg + MTX, GSK3196165 150 mg + MTX, Tofacitinib 5mg + MTX collected during the timeframe Week 0 to Week 59.
Description: The analysis was performed on the Safety Set for Pooled Placebo, GSK3196165 90 mg + MTX, GSK3196165 150 mg + MTX, Tofacitinib 5 mg + MTX. The analysis was performed on Safety Set-Period 2 for Placebo + MTX and GSK3196165 90 mg + MTX, Placebo + MTX and GSK3196165 150 mg + MTX, Placebo + MTX and Tofacitinib 5 mg + MTX.
Arm/Group | GSK3196165 90mg + MTX | GSK3196165 150mg + MTX | Tofacitinib 5mg + MTX | Pooled Placebo | Placebo + MTX and GSK3196165 90mg + MTX | Placebo + MTX and GSK3196165 150mg + MTX | Placebo + MTX and Tofacitinib 5mg + MTX
All-Cause Mortality (participants affected / at risk) | 2/513 | 7/510 | 3/273 | 1/241 | 0/80 | 1/82 | 0/68
Serious Adverse Events (participants affected / at risk) | 33/513 | 39/510 | 23/273 | 8/241 | 8/80 | 9/82 | 5/68
Other Adverse Events (participants affected / at risk) | 127/513 | 137/510 | 83/273 | 0/241 | 22/80 | 29/82 | 17/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3196165 90mg + MTX (N=513) | GSK3196165 150mg + MTX (N=510) | Tofacitinib 5mg + MTX (N=273) | Pooled Placebo (N=241) | Placebo + MTX and GSK3196165 90mg + MTX (N=80) | Placebo + MTX and GSK3196165 150mg + MTX (N=82) | Placebo + MTX and Tofacitinib 5mg + MTX (N=68)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meniere's disease (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cushing's syndrome (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Optic ischaemic neuropathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intussusception (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatorenal failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acinetobacter sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bursitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 7 (7) | 10 (10) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis staphylococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis intestinal perforated (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis E (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection pseudomonas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancoast's tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device malfunction (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conversion disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurogenic bladder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3196165 90mg + MTX (N=513) | GSK3196165 150mg + MTX (N=510) | Tofacitinib 5mg + MTX (N=273) | Pooled Placebo (N=241) | Placebo + MTX and GSK3196165 90mg + MTX (N=80) | Placebo + MTX and GSK3196165 150mg + MTX (N=82) | Placebo + MTX and Tofacitinib 5mg + MTX (N=68)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 4 (5) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 30 (54) | 35 (50) | 16 (20) | 0 (0) | 2 (2) | 2 (3) | 4 (4)
COVID-19 (Infections and infestations) | 43 (44) | 48 (48) | 29 (29) | 0 (0) | 6 (6) | 9 (9) | 2 (3)
Latent tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 3 (3) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 22 (23) | 20 (23) | 18 (22) | 0 (0) | 3 (4) | 4 (5) | 5 (6)
Urinary tract infection (Infections and infestations) | 23 (26) | 22 (26) | 19 (23) | 0 (0) | 4 (5) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 23 (29) | 31 (36) | 12 (15) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 8 (8) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-01-21): https://cdn.clinicaltrials.gov/large-docs/83/NCT03980483/Prot_002.pdf
  • Statistical Analysis Plan (2022-08-08): https://cdn.clinicaltrials.gov/large-docs/83/NCT03980483/SAP_003.pdf